Statistical Analysis Plan J2G-OX-JZJF

A Phase I, Single-Ascending Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of LOXO-292 in Healthy Adult Subjects

NCT05338515

Approval date: 03-Apr-2019



- **16.1.9 Documentation of Statistical Methods**
- 16.1.9.1 Statistical Analysis Plan

### **Statistical Analysis Plan**

A Phase I, Single-Ascending Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of LOXO-292 in Healthy Adult Subjects

Protocol No: LOXO-RET-18057 Final Protocol Date: 25 January 2019 Compound Name: LOXO-292

> Celerion Project CA27486 Final Version 1.0 Date: 03 April 2019

Loxo Oncology, Inc.
701 Gateway Boulevard, Suite 420
South San Francisco, California 94080, USA
Celerion
621 Rose Street
Lincoln, Nebraska 68502, USA
And
100 Alexis-Nihon Boulevard, Suite 360,
Montreal, QC, H4M 2N8, Canada

## Statistical Analysis Plan Signature Page

Compound Name: LOXO-292

Protocol: LOXO-RET-18057

Study Title: A Phase I, Single-Ascending Dose Study to Evaluate the Safety, Tolerability,

and Pharmacokinetics of LOXO-292 in Healthy Adult Subjects

Issue Date: 03 April 2019

| Signature: | PI<br>Date: |
|---|---|
| Pl Ph. | |
| Senior Biostatisti | cian I, Data Management and Biometrics |
| Celerion, Pi | , USA |
| PI | |
| Signature: | Date: |
| | Scientist, Clinical Pharmacology and Pharmacometrics, and Biometrics |
| Celerion, PI | , Canada |
| DocuSigned by: | |
| Signature: | Date: 03-Apr-19 13:31:39 PDT |
| PI P | Laborova this document |
| Loxo Oncology | Lapprove this document<br>3/2019 4:31:31 PM EDT<br>Inc., South San Francisco, California, USA |

## **Table of Contents**

| 1.2 | INTRODUCTION | 52 |
|---|---|---|
| 2.? | OBJECTIVES AND ENDPOINTS | 52 |
| | 2.12 Objectives | 52 |
| | 2.22 Endpoints | 52 |
| 3.2 | STUDY DESIGN | 62 |
| 4.? | ANALYSIS POPULATIONS | 72 |
| | 4.12 Analysis Populations | 72 |
| | 4.22 Preliminary Data and Interim Analysis | 72 |
| 5.2 | TREATMENT DESCRIPTIONS | 72 |
| 6.2 | PHARMACOKINETIC ANALYSIS | 82 |
| | 6.12 Measurements and Collection Schedule | 82 |
| | 6.2 Bioanalytical Method for LOXO-292 | 92 |
| | 6.32 Investigational Product and PK Analyte Information of LOXO-292 | |
| | 6.4 Pharmacokinetic Concentrations. | 92 |
| | 6.52 Noncompartmental Pharmacokinetic Analysis and Parameter Calculation for LOXO-292. | 92 |
| | 6.62 Data Summarization and Presentation | 112 |
| | 6.72 Statistical Analysis of PK Parameters | 122 |
| 7.2 | SAFETY | 132 |
| | 7.12 Subject Discontinuation | |
| | 7.22 Demographics | |
| | 7.32 Adverse Events | 142 |
| | 7.42 Clinical Laboratory Tests (Serum Chemistry, Hematology, Coagulation, and Urinalysis) | 162 |
| | 7.52 Vital Signs (Blood Pressure, Heart Rate, and Temperature) | |
| | 7.62 ECG (Heart Rate, PR, QRS, QT, and QTcF [QT with Fridericia correction]) | |
| | 7.72 Concomitant Medications | |
| | 7.82 Physical Examination | 192 |
| 8.2 | SUMMARY OF CHANGES FROM PROTOCOL-PLANNED ANALYSIS | 192 |
| 9.2 | SUMMARY TABLES AND FIGURES | 192 |
| | 9.12 In-text Summary Tables and Figures | 192 |
| | 9.2 Section 14 Summary Tables and Figures | |
| | 9.32 Section 16 Data Listings | 232 |
| 10. | TABLE AND FIGURE SHELLS | 262 |
| | 10.12 In-text Summary Tables Shells | |
| | 10.22 Figures Shells | 342 |

| Loxo Oncology, Inc. |
|---------------------------------------------|
| LOXO-292, LOXO-RET-18057 |
| Celerion, Clinical Study Report No. CA27486 |

| 10.32 Section 14 Summary Tables Shells | 44 |
|----------------------------------------|----|
| 11. TLISTING SHELLS | 63 |

#### 1. INTRODUCTION

The following statistical analysis plan (SAP) provides the framework for the summarization of the data from this study. The SAP may change due to unforeseen circumstances. Any changes made from the planned analysis within protocol, after the unblinding, or locking of the database will be documented in the clinical study report (CSR). The section referred to as Table Shells within this SAP describes the traceability of the tables, figures, and listings (TFLs) back to the data. Note that the header for this page will be the one used for the main body of the CSR.

Any additional exploratory analyses not addressed within this SAP and/or driven by the data, or requested by Loxo Oncology, Inc., will be considered out of scope and will be described in the CSR as needed.

#### 2. OBJECTIVES AND ENDPOINTS

#### 2.1 Objectives

#### Primary:

To assess the safety and tolerability of single oral doses of LOXO-292 when administered to healthy adult subjects.

#### Secondary:

To assess the PK of single oral doses of LOXO-292 when administered to healthy adult subjects.

#### 2.2 Endpoints

#### Safety:

Safety endpoints will include adverse events (AEs) including the subject incidence, number, and severity of treatment-emergent adverse events (TEAEs) following single oral doses of LOXO-292 in healthy adult subjects and safety markers for 12-lead electrocardiograms (ECGs), physical examinations, vital signs, and clinical laboratory tests.

#### **Pharmacokinetics:**

The plasma PK endpoints will include AUC0-t, AUC0-24, AUC0-inf, AUC%extrap, CL/F, Cmax, Tmax, Kel, t½, and Vz/F.

#### 3. STUDY DESIGN

This will be a Phase I, safety, tolerability, and PK single ascending dose (SAD) study. Screening of subjects will occur within 28 days prior to dosing. The study will plan to enroll up to 18 healthy, adult male and female (of non-childbearing potential only) subjects. Every attempt will be made to enroll at least 1 female in each cohort.

Up to 3 cohorts will be planned for evaluation, with 6 healthy adult subjects in each cohort. Subjects will participate in only one cohort. In each cohort, subjects will receive a single oral dose of LOXO-292 on Day 1. Cohort 2 and Cohort 3 will include a sentinel group of 2 subjects who will dose at least 48 hours before the remaining 4 subjects. Blood samples will be collected for the PK assessment of LOXO-292 in plasma for 168 hours postdose.

Safety and tolerability will be assessed through end of treatment (EOT) or early termination (ET) by monitoring AEs, performing physical examinations and clinical laboratory tests, measuring vital signs, and recording ECGs.

Dose escalation to a higher dose level (i.e., next cohort) will not take place until the Principal Investigator (PI) and Loxo Oncology, Inc. reviewed all pertinent safety and tolerability data (e.g., physical examinations, ECGs, vital signs, clinical laboratory tests, and AEs) through a minimum of 48 hours (Day 3) postdose for Cohort 1 and through a minimum of 120 hours postdose (Day 5) for Cohort 2. Following their review, the PI and Loxo Oncology, Inc. will determine that adequate safety and tolerability from the previous, lower dose, cohort had been demonstrated to permit proceeding to the next cohort. Bioanalytical data, if available, may be used to guide the dose escalation decision. Subjects may be replaced at the discretion of the Sponsor.

Subjects will be housed in the clinical research unit (CRU) from Check-in (Day -1), at the time indicated by the CRU, until after completion of the Day 8 (EOT) or ET study procedures. EOT is defined as the day on which the subject is released from the CRU, following all study procedures.

The CRUs will contact all subjects who received LOXO-292 (including subjects who terminate from the study early) at the End of Study (EOS) by a follow up (FU)phone call. The EOS/FU phone call will be performed 7 days (± 2 days) after the EOT visit or ET visit to determine if any study drug-related adverse event (AE) or serious adverse event (SAE) has occurred since the EOT or ET visit.

#### 4. ANALYSIS POPULATIONS

### 4.1 Analysis Populations

#### **Safety Population**

All subjects who received a dose of study drug will be included in the safety evaluations.

#### **Pharmacokinetic Population**

Samples from all subjects will be assayed even if the subjects do not complete the study. All subjects who comply sufficiently with the protocol and display an evaluable PK profile (e.g., exposure to treatment, availability of measurements and absence of major protocol violations) will be included in the statistical analyses. Data for each subject will be included in the summary statistics and statistical comparisons of PK parameters with the exceptions described as follows:

- Data from subjects who experience emesis at or before 2 times median Tmax for the given treatment during the PK sampling period time course of the study for LOXO-292 may be excluded from the summary statistics for the given treatment and from the statistical comparison of PK parameters.
- Data from subjects who significantly violate a protocol inclusion or exclusion criteria, deviate significantly from the protocol, or have unavailable or incomplete data that may influence the PK analysis will be excluded from the PK Population.

Any subject or data excluded from the analysis will be identified, along with the reason for exclusion, in the CSR.

All protocol deviations that occur during the study will be considered prior to database lock for their severity/impact and will be taken into consideration when subjects are assigned to analysis populations.

## 4.2 Preliminary Data and Interim Analysis

No interim analysis is planned for this study.

#### 5. TREATMENT DESCRIPTIONS

LOXO 292 will be supplied as 80 mg capsules.

All study drugs will be administered orally after an overnight fast with approximately 240 mL of water. Additional water in increments of 50 mL up to a maximum of 100 mL may be administered if needed by the subject.

Subjects will be instructed not to crush, split, or chew LOXO 292 capsules.

**Table 5.1 Treatment Descriptions** 

| Cohort | Short Description (text, tables headers, figures, listings, SAS output) | Abbreviated Description |
|---|---|---|
| 1 | 320 mg | Administration of 320 mg<br>(4 x 80 mg capsules)<br>LOXO-292 on Day 1 |
| 2 | 640 mg | Administration of 640 mg<br>(8 x 80 mg capsules)<br>LOXO-292 on Day 1 |
| 3 | 720 mg | Administration of 720 mg<br>(9 x 80 mg capsules)<br>LOXO-292 on Day 1 |

Note: additional cohorts (6 subjects per cohort) may be enrolled if it is deemed appropriate to repeat any dose level, or to add an interim dose level(s) (lower than 720 mg), as determined by Loxo Oncology, Inc in consultation with the PI, depending on the safety and tolerability results from the prior cohort(s). Dosing will not exceed 720 mg in any subject. The dose increments will be based on a review of the safety and (potentially) PK data of previous cohorts; therefore, the doses listed in this table and TFL shells are subject to change. The actual doses used in the study will be depicted in the TFLs.

#### 6. PHARMACOKINETIC ANALYSIS

#### 6.1 Measurements and Collection Schedule

Blood samples for PK assessment of LOXO-292 will be taken at the following time points on Day 1 for each cohort: predose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, 144, and 168 hours postdose.

All concentration data will be included in the calculation of the individual PK parameters, the individual concentration-time plots (based on actual sample times), and in the mean concentration-time plots (based on nominal sample times). However, if there will be any significant deviations from nominal sample times, some concentration data may be excluded from mean concentration-time plots and/or additional concentration-time plots of the mean data. All deviations and excluded data will be provided and discussed in the CSR.

## 6.2 Bioanalytical Method for LOXO-292

Plasma concentrations of LOXO-292 will be determined using a liquid chromatography-tandem mass spectrometry (LC-MS/MS) method validated with respect to accuracy, precision, linearity, sensitivity, and specificity at Alturas Analytics, Inc. (Moscow, Idaho, USA). The analytical range (lower limit of quantitation [LLOQ] – upper limit of quantitation [ULOQ]) for LOXO-292 is 1 – 1000 ng/mL. Samples that contain concentrations greater than 1000 ng/mL may be diluted up to 51-fold, if necessary, to be within the quantification range.

### 6.3 Investigational Product and PK Analyte Information of LOXO-292

LOXO-292 has a molecular weight of approximately 500 g/mol. LOXO-292 will be supplied as a powder-in-capsule containing 80 mg of drug substance (freebase) as a simple blend with excipients in a hard gelatin capsule.

#### **6.4** Pharmacokinetic Concentrations

Plasma concentrations of LOXO-292 as determined at the collection times and per the bioanalytical method described in Section 6.1 and Section 6.2, respectively, will be used for the calculation of the plasma LOXO-292 PK parameters.

# 6.5 Noncompartmental Pharmacokinetic Analysis and Parameter Calculation for LOXO-292

The appropriate noncompartmental PK parameters will be calculated from the plasma LOXO-292 concentration-time data using Phoenix® WinNonlin® Version 7.0 or higher. Actual sample times will be used in the calculations of the PK parameters. The calculation of the actual time for LOXO-292 will be in respect to the dose administration time of LOXO-292 on Day 1. All PK parameters included in the protocol are listed in Table 6.1 below, and are defined as appropriate for study design.

Table 6.1. Noncompartmental Pharmacokinetic Parameters to be Calculated for LOXO-292

| Label to be<br>Used in the<br>Text, Tables<br>and Figures | Definition | Method of<br>Determination |
|---|---|---|
| AUC0-t | Area under the concentration-time curve, from time 0 to the last observed non-zero concentration | Calculated using the Linear Trapezoidal with Linear Interpolation Method |

| Label to be<br>Used in the<br>Text, Tables | | Method of |
|---|---|---|
| and Figures | Definition | <b>Determination</b> |
| AUC0-24 | Area under the concentration-time curve from time 0 to 24 hours postdose on Day 1. If the 24-hour plasma concentration is missing, below limit of quantification (BLQ), or not reportable, then interpolation or extrapolation using the Kel will be conducted, as appropriate. If extrapolation cannot be performed, then this parameter cannot be calculated. | Calculated using the<br>Linear Trapezoidal with<br>Linear Interpolation<br>Method |
| AUC0-inf | Area under the concentration-time curve from time 0 extrapolated to infinity | Calculated as AUC0-inf = AUC0-t + (Clast/Kel) where Clast is the last observed/measured concentration |
| AUC%extrap | Percent of AUC0-inf extrapolated | Calculated as (1-AUC0-t/AUC0-inf) *100. |
| Cmax | Maximum observed concentration | Taken directly from bioanalytical data |
| Tmax | Time to reach Cmax. If the maximum value occurs at more than one time point, Tmax is defined as the first time point with this value | Taken from clinical database as the difference in the time of administration and the time of the blood draw which is associated with the Cmax. |
| Kel | Apparent terminal elimination rate constant; represents the fraction of drug eliminated per unit time | Calculated by linear least squares regression analysis using the maximum number of points in the terminal log linear phase (e.g., three or more non zero plasma concentrations). |
| t½ | Apparent first order terminal elimination half-life | Calculated as 0.693/Kel. |
| CL/F | Apparent total plasma clearance after oral (extravascular) administration | Calculated as Dose/(AUC0-inf) |
| Vz/F | Apparent volume of distribution during the terminal elimination phase after oral (extravascular) administration | Calculated as Dose/(AUC0-inf x Kel) |

Pharmacokinetic parameters will not be calculated for subjects with fewer than 3 consecutive postdose time points with quantifiable concentrations. Subjects for whom there are insufficient data to calculate the PK parameters will be included in the concentration tables only and excluded from the statistical analysis.

For the calculation of the PK parameters, plasma concentrations BLQ prior to the first quantifiable concentration will be set to 0 and plasma concentrations BLQ after the first quantifiable concentration will be treated as missing.

The Kel will be determined using linear regressions composed of least 3 data points. The Kel will not be assigned if 1) the terminal elimination phase is not apparent, 2) if Tmax is one of the 3 last data points, or 3) if the R<sup>2</sup> value is less than 0.75. In cases where the Kel interval is not assigned, the values of AUC0-inf, AUC%extrap, t½, CL/F, and Vz/F are considered not calculable and will not be reported. Wherever the resulting t½ is more than half as long as the sampling interval, the Kel values and associated parameters (AUC0-inf, AUC%extrap, t½, CL/F, and Vz/F) may not be presented as judged appropriate and in accordance with Celerion SOPs.

#### 6.6 Data Summarization and Presentation

All LOXO-292 PK concentrations and/or PK parameters descriptive statistics will be generated using SAS® Version 9.3 or higher.

The plasma concentrations of LOXO-292 will be listed and summarized by cohort and time point for all subjects in the PK Population. Plasma concentrations of LOXO-292 will be presented with the same level of precision as received from the bioanalytical laboratory. Summary statistics, including sample size (n), arithmetic mean (Mean), standard deviation (SD), coefficient of variation (CV%), standard error of the mean (SEM), minimum, median, and maximum will be calculated for all nominal concentration time points. Excluded subjects will be included in the concentration listings, but will be excluded from the summary statistics and noted as such in the tables. All BLQ values will be presented as "BLQ" in the concentration listings and footnoted accordingly.

Mean and individual concentration-time profiles will be presented on linear and semilog scales. Linear mean plots will be presented with and without SD.

Plasma LOXO-292 PK parameters will be listed and summarized by cohort for all subjects in the PK Population. Pharmacokinetic parameters will be reported to 3 significant figures for individual parameters, with the exception of Tmax, which will be presented with 2 decimal places. Summary statistics (n, arithmetic mean, SD, CV%, SEM, minimum, median, maximum, geometric mean [Geom Mean], and geometric CV% [Geom CV%]) will be calculated for plasma LOXO-292 PK parameters. Excluded subjects will be listed in the PK parameter tables, but will be excluded from the summary statistics and noted as such in the tables.

The level of precision for each concentration and PK parameter statistic will be presented as follows:

- minimum/maximum in same precision as in bioanalytical data and/or parameter output,
- mean/median in one more level of precision than minimum/maximum,
- SD/SEM in one more level of precision than mean/median,
- n will be presented as an integer,
- CV% will be presented to the nearest tenth, and
- 90% CI will be presented with 2 decimals.

## 6.7 Statistical Analysis of PK Parameters

If all three cohorts are dosed using different dose levels, dose proportionality will be evaluated graphically and using a power model. A statistical linear relationship between ln-transformed LOXO-292 parameters AUC0-t, AUC0-inf, AUC0-24, and Cmax and the ln-transformed dose will be fitted by using a regression model with ln-transformed dose as a covariate.

$$Ln(Y) = \beta_0 + \beta_1 Ln Dose + \varepsilon$$
 (Model 1)

where Y represents the PK parameter AUC0-t, AUC0-inf, AUC0-24, and Cmax.

Dose proportionality requires that  $\beta_1 = 1$  for dose-dependent parameters.

As a first step, a statistical linear relationship between the ln-transformed PK parameters AUC0-t, AUC0-inf, AUC0-24, and Cmax and the ln-transformed dose will be verified by including a quadratic (ln dose)<sup>2</sup> term in model. A 5% level of significance will be used in sequential testing of the quadratic effect. The statistical linear relationship will be concluded if the quadratic term is not statistically significant at the 0.05 probability level. If the statistical linear relationship is established in step 1, a second step will be performed. An estimate of the slope with corresponding 90% confidence interval for the quadratic term will be obtained from the power model. And, a slope around unity indicates the quadratic term is found to be supported by data; the slope near zero implies the response y is independent of (ln dose)<sup>2</sup>. If the quadratic term is not suggested from the model in the first step, the linear effect in the second step will be evaluated. In the second step, the slope of ln dose around unit suggests dose-proportionality, and the model will be used to calculate the 90% CIs for the slope of the ln-transformed PK parameters AUC0-t, AUC0-inf, AUC0-24, and Cmax.

The above assessments of dose proportionality will be performed using the following SAS® PROC MIXED code:

Step 1: To evaluate a quadratic effect:

PROC MIXED; MODEL ln(<PK Parameter>) = LDOSE LDOSE\*LDOSE / HTYPE=1; RUN;

If the quadratic term is found to be not supported by data in Step 1, and a second step will be performed to calculate the 90% CIs for the slope of the ln transformed AUC0-t, AUC0-inf, AUC0-24, and Cmax parameters. Calculation of the slope and associated 90% CI will be performed using the following SAS® PROC MIXED code:

Step 2: To evaluate a linear effect and to obtain a 90% for the slope parameter:

PROC MIXED;

MODEL LPARM = LDOSE / SOLUTION CL ALPHA=0.1 ddfm=kr outp=residuals; RUN;

Distributional assumptions underlying the statistical analyses will be assessed by visual inspection of residual plots. Normality will be examined by normal probability plots, while homogeneity of variance will be assessed by plotting the residuals against the predicted values for the model (presented in SAS output). If the assumptions are grossly violated then alternative analyses will be performed.

The following SAS code will be used to plot residuals:

PROC UNIVARIATE DATA=RESIDUALS PLOT NORMAL; VAR RESID; HISTOGRAM RESID/NORMAL; QQPLOT RESID;

If data support, plots will be provided showing individual subject values by treatment (dose) for each of the PK parameter, together with the predicted PK parameter value from the power model. For these plots, individual ln-transformed PK parameter values and ln-transformed dose values will be displayed in a scatterplot. The graph will display an estimated regression line and 90% CI. The estimated parameters of the linear regression (intercept and slope) and their 90% CIs will be included.

Dose proportionality will be concluded if a statistical linear relationship is demonstrated and if the 90% CIs around the slope estimate parameters include the value of 1 for dose dependent parameters (AUC0-t, AUC0-inf, AUC0-24, and Cmax).

#### 7. SAFETY

No inferential statistics are to be performed for the safety analysis.

All clinical safety and tolerability data will be listed by subject and assessment time points, including, unscheduled assessments (including rechecks) and early termination (ET), chronologically.

Continuous variables will be summarized using n, mean, SD, minimum, median, and maximum. Frequency counts will be reported for categorical data when appropriate.

The level of precision will be presented as follows: "n" as an integer, minimum/maximum in same precision as in the database, mean/median in one more precision level than minimum/maximum, and SD in one more precision level than mean/median.

Where individual data points are missing because of dropouts or other reasons, the data will be summarized based on reduced denominators.

When change from baseline is calculated, baseline is the last scheduled assessment before dosing in Period 1, including unscheduled assessments, whichever is later. Unscheduled assessments and ET measurements taken after first dosing will not be used in the summarization.

Note: The term 'unscheduled' assessment used in this SAP also includes recheck assessments.

### 7.1 Subject Discontinuation

Subjects will be summarized by the number of subjects enrolled, completed, and discontinued from the study with discontinuation reasons by treatment and overall. Discontinuation data will be listed by subject.

## 7.2 Demographics

Descriptive statistics will be calculated for continuous variables (age, weight, height, and body mass index) for study overall. Weight, height and body mass index are summarized at screening. Age will be derived from the date of birth to the date of dosing in Period 1. Frequency counts will be provided for categorical variables (race, ethnicity, and sex) for overall. A by-subject listing will also be provided.

#### 7.3 Adverse Events

All AEs occurring during this clinical trial will be coded using the Medical Dictionary for Regulatory Activities (MedDRA®), Version 21.1.

Each AE will be graded according to the National Institution of Health's Common Terminology Criteria for Adverse Events (CTCAE, version 5.0) using a 5-point severity scale (Grade 1, 2, 3, 4 and 5). Not all grades are appropriate for all AEs. Therefore, some AEs may be listed within the CTCAE with fewer than 5 options for grade selection.

The following clinical descriptions of severity for each AE are based on the following general guideline [CTCAE Nov2017]:

**Table 7.3: Adverse Event Severity Level and Description** 

| Grade | Description |
|---|---|
| Grade 1 | Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated. |
| Grade 2 | Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental activities of daily living (ADL)*. |
| Grade 3 | Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care ADL**. |
| Grade 4 | Life-threatening consequences; urgent intervention indicated. |
| Grade 5 | Death related to AE. |

<sup>\*</sup> Instrumental ADL refer to preparing meals, shopping for groceries or clothes, using the telephone, managing money, etc.

Similarly, the causal relationship of the study drugs to the AE will be described as Related or Unrelated to LOXO-292.

All AEs captured in the database will be listed in by-subject data listings including verbatim term, coded term, treatment group, severity grade, relationship to study drugs, and action; however, only treatment-emergent AEs (TEAEs) will be summarized.

A TEAE is defined as an undesirable event not present prior to medical treatment, or an already present event that worsens either in intensity or frequency following the treatment. Each TEAE will be attributed to a treatment based on Investigator (or designee) judgment as well as on its onset date and time. If an AE has a change in severity grade, the original AE will be given a resolution date and time of the time of severity grade increase or decrease and a new AE record will be initiated with the new severity grade, and the new AE record will use the resolved date/time of the previous record as the onset date/time. If an AE decreases in severity grade, the new AE record with less severity will be considered and counted as the same AE event of

<sup>\*\*</sup> Self-care ADL refer to bathing, dressing and undressing, feeding self, using the toilet, taking medications and not bedridden.□

the previous record with worse severity under the same treatment group in the analysis and summary tables. If the severity grade of an AE remains the same, the AE will be kept open through to resolution.

If the onset time of an AE is missing and the onset date is the same as the treatment dosing date, then the AE will be considered treatment-emergent. If the onset date of an AE is missing, then the AE will be considered treatment-emergent. If the onset date of the AE is known to have occurred prior to dosing, then the AE will not be treated as a TEAE and will instead be captured as Medical History.

TEAEs will be tabulated by system organ class and preferred term. Summary tables will include the number of subjects reporting the AE and as a percent of the number of subjects dosed by treatment and overall. Tables will also be presented by severity grade and relationship to study drugs. If a subject experienced the same TEAE more than once at a different severity grade for a given treatment, the TEAE will only be counted and presented once at the highest severity grade. Similarly, if a subject experienced the same TEAE more than once with different assessments of drug relationship for a given treatment, only the one considered related to the study drug will be counted.

Should any serious adverse events (SAEs) occur during the study, the SAEs will be displayed in a table and a narrative included in the Clinical Study Report.

# 7.4 Clinical Laboratory Tests (Serum Chemistry, Hematology, Coagulation, and Urinalysis)

All clinical laboratory test results will be presented in by-subject data listings. However, only serum chemistry, hematology, coagulation and urinalysis values will be summarized.

Hematology, coagulation, serum chemistry and urinalysis tests will be conducted at the following time points:

**Table 7.4 Lab Test Time Points** 

| Study Day |
|---------------------------------------------------|
| Screening* |
| Day -1 (check-in)* |
| Day 2** |
| Day 5 |
| Day 8** * |
| * performed following a fast of at least 12 hours |
| ** performed following a fast of at least 8 hours |
| *** performed prior to Clinic Discharge/EOT or ET |

Out-of-normal range (OOR) flags will be recorded as follows: high (H) and low (L) for numerical results and did-not-match (\*) for categorical results. If a value fails the reference range, it will automatically be compared to a computer clinically significant (CS) range suggested by the PIs (Celerion SOP GSOP.10.1028). If the value falls within the computer CS range, it will be noted as "N" for not clinically significant. If the value fails (i.e., falls outside of the CS range) the computer CS range, it will be flagged with a "Y" which prompts the PI after reviews all laboratory results to determine how the OOR value should be followed using 4 Investigator flags: "N", not clinically significant, "R", requesting a recheck, "^", checking at the next scheduled visit, or "Y", clinically significant. To distinguish the PI flag from the CS range flags, the PI flags "N" and "Y" will be presented as "-" and "+" in the data listings, respectively. Additionally, a derived flag based on a search of the PI comments for a comment of "CS" or "Clinically Significant" will be used. The derived flag will be populated with "+" if the positive clinically significant determination is found in the comments for cases when the PI flag is populated with a "^" or an "R". In addition, CTCAE, version 5.0 grading (found in NCI CTCAE guidance) will be applied to all out of range lab values deemed clinically significant by the Investigator (or designee) which are recorded as AEs.

Out-of-range values and corresponding recheck results will be listed. Other lab results within this panel and time point will also be listed for this subject. Results that are indicated as CS by the PI (either in the PI flag or in PI comments) will be listed in the table. Out-of-range values laboratory value results which are indicated as CS by PI will be reported as AEs.

For all laboratory values that are numeric, descriptive statistics (n, mean, SD, minimum, median, and maximum) will be presented for each laboratory test by treatment and time point. Change from baseline will be calculated and summarized using the Day -1 check-in value, or in the case of rechecks and unscheduled assessments the last non-missing predose measurement prior to dosing of LOXO-292. Postdose rechecks, unscheduled assessments, and ET results will not be used for calculation of descriptive statistics.

For each laboratory test, a shift table will be developed comparing the frequency of the results at baseline (above normal, normal, or below normal) to postdose results. For urinallysis tests, the categories are normal and outside normal.

All lab results, including unscheduled assessments (including rechecks), will be listed by subject.

#### 7.5 Vital Signs (Blood Pressure, Heart Rate, and Temperature)

Vital signs measurements (Blood Pressure [BP], Heart Rate [HR], and Temperature [T]) will be taken at the following time points:

**Table 7.6 Vital Signs Time Points** 

| Study Day | Study Hour | Assessment |
|---|---|---|
| Screening | | HR, HR, T <sup>†</sup> |
| Day -1 | Check-in | HR, BP, T |
| Day 1 | 0* | HR, BP, T |
| Day 1 | 2 | HR, BP |
| Day 1 | 4 | HR, BP |
| Day 1 | 24 | HR, BP |
| Day 3 | 48 | HR, BP |
| Day 4 | 72 | HR, BP |
| Day 5 | 96 | HR, BP |
| Day 6 | 120 | HR, BP |
| Day 7 | 144 | HR, BP |
| Day 8 | 168** | HR, BP, T |
| * performed within 2 hours prior dosing on Day 1 | | |
| ** performed prior to Clinic Discharge/EOT or ET | | |
| $^{\dagger}HR$ = heart rate, BP = blood pressure, T = temperature. | | |

Descriptive statistics will be reported for vital sign measurements (blood pressure and heart rate) and change from baseline by treatment and time point. Baseline is Day 1 predose value, or in the case of unscheduled assessments (including rechecks) is the last non-missing predose measurement prior to dosing. Postdose unscheduled assessments (including rechecks) and ET results will not be used for calculation of descriptive statistics. All vital signs results will be listed by subject.

## 7.6 ECG (Heart Rate, PR, QRS, QT, and QTcF [QT with Fridericia correction])

Single 12-lead ECGs measurements will be taken at the following time points:

**Table 7.7: ECG Time Points** 

| Period Day | Study Hour |
|-----------------|------------------------------------|
| Screening | |
| Day -1 | Check-in* |
| Day 1 | 3.5 (Cohorts 2 and 3 only) |
| Day 2 | 24 |
| Day 5 | 96 |
| Day 8 | 168** |
| * performed wit | hin 24 hours prior dosing on Day 1 |
| | or to Clinic Discharge/EOT or ET |

Descriptive statistics will be reported for ECG parameters and change from baseline by treatment and time point. Baseline is Day -1 check-in assessment, or in the case of

unscheduled assessments (including rechecks) is the last non-missing predose measurement prior to dosing. Postdose unscheduled assessments (including rechecks) and ET results will not be used for calculation of descriptive statistics. All ECG interval parameters will be listed by subject and time point of collection with QTcF > 450 msec and change from baseline > 30 msec flagged. All ECG results will be listed by subject.

#### 7.7 Concomitant Medications

All concomitant medications recorded during the study will be coded with the WHO Dictionary, Version 01-Sep-2018 B3 and listed.

## 7.8 Physical Examination

A full physical examination will be performed at screening and at Day 8 or upon ET. Abbreviated physical examinations will be performed at Check-in (Day -1) and 1 hour postdose. Symptom-driven physical examinations may be performed at other times, at the PI's or designee's discretion. Abnormal findings will be reported as medical history or adverse events by the clinical site. Physical examination results will be listed by subject and time point.

#### 8. SUMMARY OF CHANGES FROM PROTOCOL-PLANNED ANALYSIS

The analyses described in this SAP are aligned with those analyses described in the protocol.

#### 9. SUMMARY TABLES AND FIGURES

Summary tables and figures are numbered following the International Conference on Harmonization (ICH) structure but may be renumbered as appropriate during the compilation of the tables and figures for the CSR. Note that all summary tables and figures will be generated using SAS® Version 9.3 or higher.

## 9.1 In-text Summary Tables and Figures

The following is a list of table and figure titles that will be included in the text of the CSR. Tables and figures will be numbered appropriately during compilation of the CSR.

Section 10:

Table 10-1 Subject Disposition (Safety Population)

Section 11:

Table 11-1 Demographic Summary (Safety Population)

- Table 11-2 Summary of Plasma LOXO-292 Pharmacokinetic Parameters Following Administration of Single Ascending Doses of LOXO-292 (Cohorts 1 3) (PK Population)
- Table 11-3 Dose Proportionality Analysis of Plasma LOXO-292 Following Administration of Single Ascending Doses of LOXO-292 (Cohorts 1 3) (PK Population)
- Figure 11-1 Mean Plasma LOXO-292 Concentrations-Time Profiles Following Administration of a Single Dose of LOXO-292 (Cohorts 1 3) (Linear Scale) (PK Population)
- Figure 11-2 Dose Proportionality of Plasma LOXO-292 AUC0-t Following Administration of Single Ascending Doses of LOXO-292 (PK Population) (Log Scale)
- Figure 11-3 Dose Proportionality of Plasma LOXO-292 AUC0-24 Following Administration of Single Ascending Doses of LOXO-292 (PK Population) (Log Scale)
- Figure 11-4 Dose Proportionality of Plasma LOXO-292 AUC0-inf Following Administration of Single Ascending Doses of LOXO-292 (PK Population) (Log Scale)
- Figure 11-5 Dose Proportionality of Plasma LOXO-292 Cmax Following Administration of Single Ascending Doses of LOXO-292 (PK Population) (Log Scale)

#### Section 12:

Table 12-1 Adverse Event Frequency by Treatment - Number of Subjects Reporting the Event (% of Subjects Dosed)

## 9.2 Section 14 Summary Tables and Figures

The following is a list of table and figure titles that will be included in Section 14 of the report. Table and figure titles may be renumbered as appropriate during the compilation of the report.

#### 14.1 Demographic Data Summary Tables

- Table 14.1.1 Summary of Disposition (Safety Population)
- Table 14.1.2 Disposition of Subjects (Safety Population)
- Table 14.1.3 Demographic Summary (Safety Population)

#### 14.2 Pharmacokinetic Data Summary Tables and Figures

## 14.2.1 Plasma LOXO-292 Tables

- Table 14.2.1.1 Plasma LOXO-292 Concentrations (ng/mL) Following Administration of a Single Oral Dose of 320 mg LOXO-292 (Cohort 1) (PK Population)
- Table 14.2.1.2 Plasma LOXO-292 Concentrations (ng/mL) Following Administration of a Single Dose of 640 mg LOXO-292 (Cohort 2) (PK Population)
- Table 14.2.1.3 Plasma LOXO-292 Concentrations (ng/mL) Following Administration of a Single Dose of 720 mg LOXO-292 (Cohort 3) (PK Population)
- Table 14.2.1.4 Plasma LOXO-292 Pharmacokinetic Parameters Following Administration of a Single Dose of 320 mg LOXO-292 (Cohort 1) (PK Population)
- Table 14.2.1.5 Plasma LOXO-292 Pharmacokinetic Parameters Following Administration of a Single Dose of 640 mg LOXO-292 (Cohort 2) (PK Population)
- Table 14.2.1.6 Plasma LOXO-292 Pharmacokinetic Parameters Following Administration of a Single Dose of 720 mg LOXO-292 (Cohort 3) (PK Population)
- Table 14.2.1.7 Intervals (Hours) Used for Determination of Plasma LOXO-292 Kel Values Following Administration of a Single Dose of LOXO-292 (Cohorts 1 3) (PK Population)
- Table 14.2.1.8 Dose Proportionality Analysis of Plasma LOXO-292 Following Administration of Single Ascending Doses of LOXO-292 (Cohorts 1 3) (PK Population)

## 14.2.2 Plasma LOXO-292 Figures

- Figure 14.2.2.1 Mean (SD) Plasma LOXO-292 Concentration-Time Profiles Following Administration of Single Ascending Doses of LOXO-292 (Linear Scale) (PK Population)
- Figure 14.2.2.2 Mean Plasma LOXO-292 Concentration-Time Profiles
  Following Administration of Single Ascending Doses of
  LOXO-292 (Linear Scale) (PK Population)
- Figure 14.2.2.3 Mean Plasma LOXO-292 Concentration-Time Profiles Following Administration of Single Ascending Doses of LOXO-292 (Semi-Log Scale) (PK Population)
- Figure 14.2.2.4 Dose Proportionality of Plasma LOXO-292 AUC0-t Following Administration of Single Ascending Doses of LOXO-292 (PK Population) (Log Scale)

- Figure 14.2.2.5 Dose Proportionality of Plasma LOXO-292 AUC0-24 Following Administration of Single Ascending Doses of LOXO-292 (PK Population) (Log Scale)
- Figure 14.2.2.6 Dose Proportionality of Plasma LOXO-292 AUC0-inf Following Administration of Single Ascending Doses of LOXO-292 (PK Population) (Log Scale)
- Figure 14.2.2.7 Dose Proportionality of Plasma LOXO-292 Cmax Following Administration of Single Ascending Doses of LOXO-292 (PK Population) (Log Scale)

## 14.3 Safety Data Summary Tables

## 14.3.1 Displays of Adverse Events

- Table 14.3.1.1 Treatment-emergent Adverse Event Frequency by Treatment
   Number of Subjects Reporting Events (% of Subject
  Dosed) (Safety Population)
- Table 14.3.1.2 Treatment-Emergent Adverse Event Frequency by
  Treatment, Severity Grade, and Relationship to Study Drugs
   Number of Subjects Reporting Events (Safety Population)

### 14.3.2 Listings of Deaths, other Serious and Significant Adverse Events

Table 14.3.2.1 Serious Adverse Events (Safety Population)

<If no serious adverse event occurred, a statement 'There was no serious adverse event recorded during the study.' will be added.>

# 14.3.3 Narratives of Deaths, other Serious and Certain other Significant Adverse Events

#### 14.3.4 Abnormal Laboratory Value Listing (each patient)

- Table 14.3.4.1 Out-of-Range Values and Recheck Results Serum Chemistry (Safety Population)
- Table 14.3.4.2 Out-of-Range Values and Recheck Results Hematology and Coagulation
- Table 14.3.4.3 Out-of-Range Values and Recheck Results Urinalysis
- Table 14.3.4.4 Clinically Significant Laboratory and Corresponding Results (Safety Population)

# 14.3.5 Displays of Other Laboratory, Vital Signs, Electrocardiogram, Physical Examination, and Other Safety Data

Table 14.3.5.1 Clinical Laboratory Summary and Change from Baseline – Serum Chemistry (Safety Population)

| Table 14.3.5.2 | Clinical Laboratory Shift from Baseline – Serum Chemistry (Safety Population) |
|---|---|
| Table 14.3.5.3 | Clinical Laboratory Summary and Change from Baseline – Hematology (Safety Population) |
| Table 14.3.5.4 | Clinical Laboratory Shift from Baseline – Hematology (Safety Population) |
| Table 14.3.5.5 | Clinical Laboratory Summary and Change from Baseline – Urinalysis (Safety Population) |
| Table 14.3.5.6 | Clinical Laboratory Shift from Baseline – Urinalysis (Safety Population) |
| Table 14.3.5.7 | Vital Sign Summary and Change from Baseline (Safety Population) |
| Table 14.3.5.8 | 12-Lead Electrocardiogram Summary and Change from Baseline (Safety Population) |

## 9.3 Section 16 Data Listings

Note: Virology test results (Hepatitis and HIV) that are provided by the clinical laboratory will not be presented in subject data listings and will not be included in the database transfer.

Data listings are numbered following the ICH structure but may be renumbered as appropriate during the compilation of the TFLs for the CSR. The following is a list of appendix numbers and titles that will be included as data listings:

#### **16.1** Study Information

Appendix 16.1.9 Statistical Methods

Appendix 16.1.10.1 Clinical Laboratory Reference Ranges

## 16.2 Subject Data Listings

### **16.2.1** Subject Discontinuation

Appendix 16.2.1 Subject Discontinuation (Safety Population)

#### **16.2.2** Protocol Deviations

Appendix 16.2.2 Protocol Deviations

# 16.2.3 Subjects Excluded from < Pharmacokinetic/Efficacy > Analysis

Appendix 16.2.3 Subjects Excluded from < Pharmacokinetic/Efficacy> Analysis

<Note: Appendices 16.2.2 and 16.2.3 are generated in MS Word for inclusion in the study report.>

# 16.2.4 Demographic Data

| Appendix 16.2.4.1 | Demographics (Safety Population) |
|-------------------|--------------------------------------------------|
| Appendix 16.2.4.2 | Updated Informed Consent (Safety Population) |
| Appendix 16.2.4.3 | Physical Examination (Safety Population) |
| Appendix 16.2.4.4 | Medical and Surgical History (Safety Population) |

## 16.2.5 Compliance and/or Drug Concentration Data

| Appendix 16.2.5.1.1 | Inclusion Criteria |
|---------------------|--------------------------------------------------------|
| Appendix 16.2.5.1.2 | Exclusion Criteria |
| Appendix 16.2.5.2 | Subject Eligibility (Safety Population) |
| Appendix 16.2.5.3 | Check-in Criteria and Responses (Safety Population) |
| Appendix 16.2.5.4.1 | Test Compound Description (Safety Population) |
| Appendix 16.2.5.4.2 | Test Compound Administration Times (Safety Population) |
| Appendix 16.2.5.5 | Blood Draw Times (Safety Population) |
| Appendix 16.2.5.6 | Meal Times (Safety Population) |
| Appendix 16.2.5.7 | Concomitant Medications (Safety Population) |

## 16.2.6 Individual Pharmacokinetic Response Data

| Appendix 16.2.6.1 | Individual Plasma LOXO-292 Concentrations Versus Time Profiles Following Administration of a Single Dose of 320 mg LOXO-292 for Subject X (Cohort 1) (Linear and Semi-Log Scale) |
|---|---|
| Appendix 16.2.6.2 | Individual Plasma LOXO-292 Concentrations Versus Time Profiles Following Administration of a Single Dose of 640 mg LOXO-292 for Subject X (Cohort 2) (Linear and Semi-Log Scale) |

| Appendix 16.2.6.3 | Individual Plasma LOXO-292 Concentrations Versus |
|-------------------|----------------------------------------------------|
| | Time Profiles Following Administration of a Single |
| | Dose of 720 mg LOXO-292 for Subject X (Cohort 3) |
| | (Linear and Semi-Log Scale) |

# **16.2.7** Adverse Events Listings

| Appendix 16.2.7.1 | Adverse Events (I of II) (Safety Population) |
|---|---|
| Appendix 16.2.7.2 | Adverse Events (II of II) (Safety Population) |
| Appendix 16.2.7.3 | Adverse Event Non-Drug Therapy (Safety Population) |
| Appendix 16.2.7.4 | Adverse Event Preferred Term Classification (Safety Population) |

# 16.2.8 Listings of Individual Laboratory Measurements and Other Safety Observations

| Appendix 16.2.8.1.1 | Clinical Laboratory Report - Serum Chemistry (Safety Population) |
|---|---|
| Appendix 16.2.8.1.2 | Clinical Laboratory Report - Hematology (Safety Population) |
| Appendix 16.2.8.1.3 | Clinical Laboratory Report - Urinalysis (Safety Population) |
| Appendix 16.2.8.1.4 | Clinical Laboratory Report - Urine Drug Screening (Safety Population) |
| Appendix 16.2.8.1.5 | Clinical Laboratory Report - Other (Safety Population) |
| Appendix 16.2.8.1.6 | Clinical Laboratory Report - Comments (Safety Population) |
| Appendix 16.2.8.2 | Vital Signs (Safety Population) |
| Appendix 16.2.8.3 | 12-Lead Electrocardiogram (Safety Population) |
| Appendix 16.2.8.4 | Phone Call (Safety Population) |

#### 10. TABLE AND FIGURE SHELLS

The following table shells provide a framework for the display of data from this study. The shells may change due to unforeseen circumstances. These shells may not be reflective of every aspect of this study, but are intended to show the general layout of the tables and figures that will be presented and included in the final CSR. Unless otherwise noted, all in-text tables will be presented in Times New Roman font size 8 and post-text tables in Courier New size font 9. These tables will be generated according to the ADaM Model 2.1 and ADaM implementation guide 1.1.

# 10.1 In-text Summary Tables Shells

Table 10-1 Summary of Disposition (Safety Population)

| Disposition | 320 mg | 640 mg | 720 mg | Overall |
|---------------------|-----------|-----------|-----------|-----------|
| Enrolled | XX (100%) | XX (100%) | XX (100%) | XX (100%) |
| Completed Study | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) |
| Discontinued Early | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) |
| <reason1></reason1> | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) |
| <reason2></reason2> | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) |

320 mg LOXO-292: Administration of 320 mg (4 x 80 mg capsules) LOXO-292 on Day 1

640 mg LOXO-292: Administration of 320 mg (8 x 80 mg capsules) LOXO-292 on Day 1

720 mg LOXO-292: Administration of 320 mg (9 x 80 mg capsules) LOXO-292 on Day 1

Source: Table 14.1.1.1

Program: /CAXXXXX/sas\_prg/stsas/intext/t\_disp.sas\_DDMMMYYYY HH:MM

Table 11-1 Demographic Summary (Safety Population)

| Trait | | 320 mg | 640 mg | 720 mg | Study Overall |
|---|---|---|---|---|---|
| Sex | Male | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) |
| | Female | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) |
| Race | Asian | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) |
| | Black or African<br>American | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) |
| | White | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) |
| Ethnicity | Hispanic or Latino | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) |
| | Not Hispanic or Latino | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) |
| Age* (yr) | n | XX | XX | XX | XX |
| | Mean | XX.XX | XX.XX | XX.XX | XX.XX |
| | SD | XX.XXX | XX.XXX | XX.XXX | XX.XXX |
| | Minimum | XX.XX | XX.XX | XX.XX | XX.XX |
| | Median | XX.X | XX.X | XX.X | XX.X |
| | Maximum | XX.XX | XX.XX | XX.XX | XX.XX |
| Height (cm) | n | XX | XX | XX | XX |
| | Mean | XXX.X | XXX.X | XXX.X | XXX.X |
| | SD | X.XX | X.XX | X.XX | X.XX |
| | Minimum | XXX | XXX | XXX | XXX |
| | Median | XXX.X | XXX.X | XXX.X | XXX.X |
| | Maximum | XXX | XXX | XXX | XXX |

320 mg LOXO-292: Administration of 320 mg (4 x 80 mg capsules) LOXO-292 on Day 1

640 mg LOXO-292: Administration of 320 mg (8 x 80 mg capsules) LOXO-292 on Day 1

BMI = Body mass index

Source: Table 14.1.1.3

Program: /CAXXXXX/sas\_prg/stsas/intexttest/t\_dem.sas DDMMMYYYY HH:MM

**Programmer Note:** Weight (kg) and BMI (kg/m²) will also be summarized in the table above.

<sup>720</sup> mg LOXO-292: Administration of 320 mg (9 x 80 mg capsules) LOXO-292 on Day 1

<sup>\*</sup> Age is calculated from the date of first dosing.

## Table 11-2 will be in the following format:

Table 11-2 Summary of Plasma LOXO-292 Pharmacokinetic Parameters Following Administration of Single Ascending Doses of LOXO-292 (Cohorts 1 – 3) (PK Population)

| Pharmacokinetic<br>Parameters | 320 mg | 640 mg | 720 mg |
|---|---|---|---|
| Param1 (units) | XXX.X (XX.X) [n=xx] | XXX.X (XX.X) [n=xx] | XXX.X (XX.X) [n=xx] |
| Param2 (units) | XXX.X (XX.X) [n=xx] | XXX.X (XX.X) [n=xx] | XXX.X (XX.X) [n=xx] |
| Param3 (units) | XXX.X (XX.X) [n=xx] | XXX.X (XX.X) [n=xx] | XXX.X (XX.X) [n=xx] |
| Param4 (units) | XXX.X (XX.X) [n=xx] | XXX.X (XX.X) [n=xx] | XXX.X (XX.X) [n=xx] |

320 mg LOXO-292: Administration of 320 mg (4 x 80 mg capsules) LOXO-292 on Day 1

640 mg LOXO-292: Administration of 320 mg (8 x 80 mg capsules) LOXO-292 on Day 1

720 mg LOXO-292: Administration of 320 mg (9 x 80 mg capsules) LOXO-292 on Day 1

AUCs and Cmax values are presented as geometric mean and geometric CV%.

Tmax values are presented as median (min, max).

Other parameters are presented as arithmetic mean  $(\pm SD)$ .

Source: Tables 14.2.1.4 through 14.2.1.6

#### Notes for Generating the Actual Table:

Presentation of Data:

- The following PK parameters will be presented in the following order and with following units: AUCO-24 (ng\*hr/mL), AUCO-t (ng\*hr/mL), AUCO-t (ng\*hr/mL), AUCO-t (ng\*hr/mL), AUCO-t (ng\*hr/mL), Tmax (hr), Kel (1/hr), t½ (hr), CL/F (L/hr), and Vz/F (L)
- n will be presented as an integer (with no decimal);
- · Summary statistics will be presented with same precision as defined in post-text shells

Celerion Note: Per study design needs, the following changes are made to this table relative to Celerion's standard shell:

1. Add the third treatment column to this table and update title

Program: /CAXXXXX/sas\_prg/pksas/intext-pk-tables.sas DDMMYYYY HH:MM
Program: /CAXXXXX/sas\_prg/pksas/adam\_intext\_pkparam.sas DDMMYYYY HH:MM

Table 11-3 will be in the following format:

Table 11-3 Dose Proportionality Analysis of Plasma LOXO-292 Following Administration of Single Ascending Doses of LOXO-292 (Cohorts 1 – 3) (PK Population)

| Pharmacokinetic<br>Parameters | Estimate of Slope (b) | Standard error | 90% Confidence Interval for Slope |
|---|---|---|---|
| param1 | X.XXXX | X.XXXX | X.XXXX - X.XXXX |
| param2 | X.XXXX | X.XXXX | X.XXXX - X.XXXX |
| param3 | X.XXXX | X.XXXX | X.XXXX - X.XXXX |
| param4 | X.XXXX | X.XXXX | X.XXXX - X.XXXX |

Parameters were In-transformed prior to analysis.

The following statistical model using PROC MIXED of SAS was used to test dose proportionality:

Parameter =  $a * Dose^b$  which was equivalent to ln(Parameter) = ln(a) + b[ln(Dose)]

Dose proportionality is not rejected if the 90% CI for b contains 1.

Source: Table 14.2.1.6

## Notes for Generating the Actual Table:

PK Parameters are AUCO-24, AUCO-t, AUCO-inf, and Cmax

Please use the footnote below:

Parameters were In-transformed prior to analysis.

The following statistical model using PROC MIXED of SAS was used to test dose proportionality: Parameter =  $a * Dose^b$  which was equivalent to ln(Parameter) = ln(a) + b[ln(Dose)]

Dose proportionality is not rejected if the 90% CI for b contains 1.

#### Presentation of Data:

- · Slope will be presented to 4 decimal places
- · Standard error will be presented to 4 decimal places
- 90% CI will be presented to 4 decimal places

Program: /CAXXXXX/sas\_prg/pksas/doseprop-mixed.sas DDMMMYYYY HH:MM

Table 12-1 Treatment-Emergent Adverse Event Frequency by Treatment –
Number of Subjects Reporting the Event (% of Subjects Dosed) (Safety Population)

| Adverse Events* | 320 mg | 640 mg | 720 mg | Overall |
|---|---|---|---|---|
| Number of Subjects Dosed | XX (100%) | XX (100%) | XX (100%) | XX (100%) |
| Number of Subjects With TEAEs | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) |
| Number of Subjects Without TEAEs | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) |
| System Organ Class 1 | X (X%) | X ( X%) | X ( X%) | X (X%) |
| Preferred Term 1 | X (X%) | X (X%) | X (X%) | X ( X%) |
| Preferred Term 2 | X (X%) | X (X%) | X ( X%) | X (X%) |
| System Organ Class 2 | X (X%) | X (X%) | X (X%) | X ( X%) |
| Preferred Term 1 | X (X%) | X (X%) | X ( X%) | X (X%) |
| Preferred Term 2 | X (X%) | X (X%) | X ( X%) | X (X%) |

320 mg LOXO-292: Administration of 320 mg (4 x 80 mg capsules) LOXO-292 on Day 1

640 mg LOXO-292: Administration of 320 mg (8 x 80 mg capsules) LOXO-292 on Day 1

Although a subject may have had 2 or more clinical adverse experiences, the subject is counted only once within a category. The same subject may appear in different categories.

For an AE with multiple changes in severity, a new record with severity less or equal to its maximum severity will not be included in the adverse event summary tables.

Source: Table 14.3.1.1

Program: /CAXXXXX/sas prg/stsas/intexttest/t ae.sas DDMMMYYYY HH:MM

Programmer Note: Sort by decreasing frequency of system organ class and by preferred term within a system organ class of Overall column.

<sup>720</sup> mg LOXO-292: Administration of 320 mg (9 x 80 mg capsules) LOXO-292 on Day 1

<sup>\*</sup> Adverse events are coded using MedDRA® Version 21.1 by System Organ Class and Preferred Term.

TEAE = Treatment-emergent Adverse event

## 10.2 Figures Shells

Figures 11-1 and 14.2.2.2 will be in the following format:

Figure 11-1 Mean Plasma LOXO-292 Concentrations-Time Profiles Following Administration of Single Ascending Doses of LOXO-292 (Cohorts 1 – 3) (Linear Scale) (PK Population)



Program: /CAXXXXX/sas\_prg/pksas/adam\_meangraph.sas DDMMMYYY HH:MM Program: /CAXXXXX/sas\_prg/pksas/meangraph.sas DDMMMYYY HH:MM
# Notes for Generating the Actual Mean Figure:

- Legend will be "320 mg LOXO-292", "640 mg LOXO-292", and "720 mg LOXO-292"
- Y axis label will be "Plasma LOXO-292 Concentration (ng/mL)"
- X axis label will be "Time (hr)"
- Add in footnote: LLOQ value for LOXO-292 in plasma is 1.00 ng/mL

Program: /CAXXXX/sas\_prg/pksas/meangraph.sas DDMMMYYYY HH:MM

Program: /CAXXXXX/sas\_prg/pksas/adam\_meangraph.sas DDMMMYYYYY HH:MM

Figure 14.2.2.1 will be in the following format:

Figure 14.2.2.1 Mean (SD) Plasma LOXO-292 Concentration-Time Profiles Following Administration of Single Ascending Doses of LOXO-292 (Linear Scale) (PK Population)



Treatments B and C are shifted to the right for ease of reading

 $Program: \ /CAXXXXX/sas\_prg/pksas/adam\_meangraph.sas \ DDMMMYYY \ HH:MM$ 

Program: /CAXXXXX/sas prg/pksas/meangraph.sas DDMMMYYY HH:MM

# Notes for Generating the Actual Mean Figure:

- Legend will be "320 mg LOXO-292", "640 mg LOXO-292", and "720 mg LOXO-292"
- Y axis label will be "Plasma LOXO-292 Concentration (ng/mL)"
- X axis label will be "Time (hr)"
- Add the following footnote: "640 mg LOXO-292 and 720 mg LOXO-292 are shifted to the right for ease of reading"
- Add in footnote: LLOQ value for LOXO-292 in plasma is 1.00 ng/mL

Program: /CAXXXX/sas\_prg/pksas/meangraph.sas DDMMMYYYY HH:MM

Program: /CAXXXXX/sas\_prg/pksas/adam\_meangraph.sas DDMMMYYYY HH:MM

Figure 14.2.2.3 will be in the following format:

Figure 14.2.2.3 Mean Plasma LOXO-292 Concentration-Time Profiles Following Administration of Single Ascending Doses of LOXO-292 (Semi-Log Scale) (PK Population)



Program: /CAXXXXX/sas\_prg/pksas/adam\_meangraph.sas DDMMMYYY HH:MM Program: /CAXXXXX/sas\_prg/pksas/meangraph.sas DDMMMYYY HH:MM

# Notes for Generating the Actual Mean Figure:

- Legend will be "320 mg LOXO-292", "640 mg LOXO-292", and "720 mg LOXO-292"
- Y axis label will be "Plasma LOXO-292 Concentration (ng/mL)"
- X axis label will be "Time (hr)"
- Add in footnote: LLOQ value for LOXO-292 in plasma is 1.00 ng/mL

Program: /CAXXXXX/sas\_prg/pksas/meangraph.sas DDMMMYYYY HH:MM

Program: /CAXXXXX/sas\_prg/pksas/adam\_meangraph.sas DDMMMYYYYY HH:MM

Figures 11-2 through 11-5 and 14.2.2.4 through 14.2.2.7 will be in the following format:

Figure 11-2 Dose Proportionality of Plasma LOXO-292 AUC0-t Following Administration of Single Ascending Doses of LOXO-292 (PK Population) (Log Scale)

\*\*\* Note: this is not a Celerion standard figure \*\*\*

# Notes for Generating the Actual Mean Figure:

- Legend will be "320 mg LOXO-292", "640 mg LOXO-292", and "720 mg LOXO-292"
- Y axis label will be "AUCO-24 (ng\*hr/mL), AUCO-t (ng\*hr/mL), AUCO-inf (ng\*hr/mL), and Cmax (ng/mL)" as appropriate (Log scale)
- X axis will be "LOXO-292 Dose (mg)" (Log scale)

Appendix 16.2.6.1

Individual Plasma LOXO-292 Concentration-Time Profiles Following Administration of a Single Dose of 320 mg LOXO-292 for Subject X (Cohort 1) (Linear and Semi-Log Scale)



Program: /CAXXXXX/sas\_prg/pksas/adam\_indgraph.sas DDMMMYYY HH:MM Program: /CAXXXXX/sas\_prg/pksas/indgraph-all.sas DDMMMYYY HH:MM

### Notes for Generating the Actual Individual Figure:

- Use same format for Appendix 16.2.6.1 through 16.2.6.3
- Legend will be "320 mg LOXO-292" for Appendix 16.2.6.1
- Legend will be "640 mg LOXO-292" for Appendix 16.2.6.2
- Legend will be "720 mg LOXO-292" for Appendix 16.2.6.3
- Y axis label will be "Plasma LOXO-292 Concentration (ng/mL)"
- X axis label will be "Hours"
- Add in footnote: LLOQ value for LOXO-292 in plasma is 1.00 ng/mL

Program: /CAXXXXX/sas\_prg/pksas/indgraph-all.sas DDMMMYYYY HH:MM Program: /CAXXXXX/sas\_prg/pksas/adam\_indgraph.sas DDMMMYYYY HH:MM

# 10.3 Section 14 Summary Tables Shells

Page X of X

Table 14.1.1 Summary of Disposition (Safety Population)

| Disposition | 320 mg | 640 mg | 720 mg | Overall |
|--------------------|--------|--------|--------|---------|
| Enrolled | X | X | X | XX |
| Completed | X | X | X | XX |
| Discontinued Early | X | X | X | XX |
| Reason 1 | X | X | X | XX |
| Reason 2 | X | X | X | XX |
| Reason 3 etc. | Х | Х | Х | XX |

Note: 320 mg: Administration of 320 mg (4 x 80 mg capsules) LOXO-292 on Day 1  $\,$ 

640 mg: Administration of 320 mg (8 x 80 mg capsules) LOXO-292 on Day 1

720 mg: Administration of 320 mg (9 x 80 mg capsules) LOXO-292 on Day 1  $\,$ 

Table 14.1.2 Disposition of Subjects (Safety Population)

| Subject | | | | Study Completion | |
|---|---|---|---|---|---|
| Number | Treatment | Dosed | Completed | Status | Date |
| XXX-XXX<br>XXX-XXX | XXX mg | Yes<br>Yes | Yes<br>No | Completed Study<br>Withdrew Consent | DDMMYYYY<br>DDMMYYYY |

Note: 320 mg: Administration of 320 mg (4  $\times$  80 mg capsules) LOXO-292 on Day 1 640 mg: Administration of 320 mg (8  $\times$  80 mg capsules) LOXO-292 on Day 1 720 mg: Administration of 320 mg (9  $\times$  80 mg capsules) LOXO-292 on Day 1

Table 14.1.3 Demographic Summary (Safety Population)

| Trait | | 320 mg | 640 mg | 720 mg | Study<br>Overall |
|---|---|---|---|---|---|
| Sex | Male | X ( XX%) | X ( XX%) | X ( XX%) | X ( XX%) |
| | Female | X ( XX%) | X ( XX%) | X ( XX%) | X ( XX%) |
| Race | Asian | X ( XX%) | X (XX%) | X ( XX%) | X (XX%) |
| | Black or African American | X ( XX%) | X ( XX%) | X ( XX%) | X ( XX%) |
| | White | X ( XX%) | X ( XX%) | X ( XX%) | X ( XX%) |
| Ethnicity | Hispanic or Latino | X ( XX%) | X (XX%) | X (XX%) | X (XX%) |
| | Not Hispanic or Latino | X ( XX%) | X ( XX%) | X ( XX%) | X ( XX%) |
| Age*(yr) | n | XX | XX | XX | XX |
| 50 NEW 97. | Mean | XX.X | XX.X | XX.X | XX.X |
| | SD | X.XX | X.XX | X.XX | X.XX |
| | Minimum | XX | XX | XX | XX |
| | Median | XX.X | XX.X | XX.X | XX.X |
| | Maximum | XX | XX | XX | XX |
| Height (cm) | n | XX | XX | XX | XX |
| Accessors - Marie Accessors | Mean | XX.X | XX.X | XX.X | XX.X |
| | SD | X.XX | X.XX | X.XX | X.XX |
| | Minimum | XX | XX | XX | XX |
| | Median | XX.X | XX.X | XX.X | XX.X |
| | Maximum | XX | XX | XX | XX |

Programmer Note: Also include weight (kg) and BMI (kg/m²)

Note: \* Age is calculated from the date of first dosing.

BMI = Body mass index

320 mg: Administration of 320 mg (4 x 80 mg capsules) LOXO-292 on Day 1

640 mg: Administration of 320 mg (8 x 80 mg capsules) LOXO-292 on Day 1

720 mg: Administration of 320 mg (9 x 80 mg capsules) LOXO-292 on Day 1

# Tables 14.2.1.1 through 14.2.1.3 will be in the following format:

Table 14.2.1.1 Plasma LOXO-292 Concentrations (ng/mL) Following Administration of a Single Dose of 320 mg LOXO-292 (Cohort 1) (PK Population)

| Subject | Sample Times (hr) | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Number | Predose | XX | XX | XX | XX | XX | XX | XX | XX |
| X | BLQ | XX | XX | XX | XX | XX | XX | XX | XX |
| X | BLQ | XX | XX | XX | XX | XX | XX | XX | XX |
| X | BLQ | XX | XX | XX | XX | XX | XX | XX | XX |
| n | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| CV% | | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SEM | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Minimum | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Maximum | XX | XX | XX | XX | XX | XX | XX | XX | XX |

For the calculation of summary statistics, values that are below the limit of quantitation (BLQ) of 1 ng/mL are treated as 0 before the first quantifiable concentration and as missing elsewhere.

<sup>. =</sup> Value missing or not reportable.

### Notes for Generating the Actual Table:

Presentation of Data:

Concentrations will be presented to same precision as in bio data.

Summary statistics presentation with respect to the precision of the bio data: n = integer; Mean and Median +1; SD and SEM +2, Min and Max +0, CV% to 1 decimal

DDMMMYYYY HH:MM

Programmer Note:

PK Time points are: predose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, 144, and 168 hours postdose.

#### Per study design needs, the following changes are made to this table relative to Celerion standard:

1. Please remove the <Treatment Sequence> and <Study Period> columns from all tables.

| Program: | milling pk-conc-tables-sig.sas | DDMMYYYYY | HH:MM |
|----------|-----------------------------------------|-----------|-------|
| | 100000000000000000000000000000000000000 | | |
| ] | | | |
| 1 | | | |

# Tables 14.2.1.4 through 14.2.1.6 will be in the following format:

Table 14.2.1.4 Plasma LOXO-292 Pharmacokinetic Parameters Following Administration of a Single Dose of 320 mg LOXO-292 (Cohort 1) (PK Population)

| | | | F | arameters | | |
|-----------|---------|---------|---------|-----------|---------|---------|
| Subject | param1 | param2 | param3 | param4 | param5 | param6 |
| Number | (units) | (units) | (units) | (units) | (units) | (units) |
| X | XXX | X.XX | XXX | XXX | XX.X | X.XXX |
| X | XX.X | X.XX | XXX | XXX | XX.X | X.XXX |
| X | XXX | X.XX | XXX | XXX | XX.X | X.XXX |
| X | XX.X | X.XX | XXX | XXX | XX.X | X.XXX |
| X | XX.X | X.XX | XXX | XXX | XX.X | X.XXX |
| X | X.XX | X.XX | XXX | XXX | XX.X | X.XXX |
| X | XXX | X.XX | XXX | XXX | XX.X | X.XXX |
| n | XX | XX | XX | XX | XX | XX |
| Mean | XXX.X | X.XXX | XXX.X | XXX.X | XX.XX | X.XXXX |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| CV% | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SEM | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Minimum | XX.X | X.XX | XXX | XXX | XX.X | X.XXX |
| Median | XX.XX | X.XXX | XXX.X | XXX.X | XX.XX | X.XXXX |
| Maximum | XXX | X.XX | XXX | XXX | XX.X | X.XXX |
| Geom Mean | XXX.X | X.XXX | XXX.X | XXX.X | XX.XX | X.XXXX |
| Geom CV% | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |

-----

<sup>. =</sup> Value missing or not reportable.

#### Notes for Generating the Actual Table:

#### Presentation of Data:

- PK Parameters will be presented in the following order and with following units: AUCO-24 (ng\*hr/mL), AUCO-t (ng\*hr/mL), AUCO-inf (ng\*hr/mL), AUC%extrap (%), Cmax (ng/mL), Tmax (hr), Kel (1/hr), t1/2 (hr), CL/F (L/hr), and Vz/F (L)
- n will be presented as an integer (with no decimal);
- Parameter values for exposure based parameters (i.e. AUCs, Cmax, Vz/F, and CL/F) will be presented with, at maximum, the precision of the bio data, and, at minimum, 3 significant figures (to be determined by the PKist once bio data are received). Summary statistics for exposure parameters will be presented as: Mean, Median, and Geom Mean+1; SD and SEM +2, Min and Max +0.
- Values for time-based parameters (i.e. Tmax and t1/2) will be presented with 2 decimals. Summary statistics for time-based parameters will be presented as: Mean, Median, and Geom Mean +1; SD +2, Min and Max +0.
- Values for rate constants (i.e. Kel) will be presented with 3 significant figures. Summary statistics for Kel will be presented as: Mean, Median, and Geom Mean +1; SD and SEM +2, Min and Max +0.
- . CV% and Geom CV% for all parameters will be presented with 1 decimal

#### Per study design needs, the following changes are made to this table relative to Celerion standard:

1. Please remove the "Treatment Sequence" and "Study Period" columns.

Program: /CAXXXX/sas\_prg/pksas/pk-tables.sas DDMMMYYYY HH:MM

Program: /CAXXXXX/sas\_prg/pksas/adam\_pkparam.sas DDMMMYYYY HH:MM

### Table 14.2.1.7 will be in the following format:

Table 14.2.1.7 Intervals (Hours) Used for Determination of Plasma LOXO-292 Kel Values Following Administration of a Single Dose of LOXO-292 (Cohorts 1 - 3) (PK Population)

| Subject<br>Number | Treatment | Interval | R2 | n |
|-------------------|-----------|-------------|-------|---|
| Х | Х | xx.x - xx.x | x.xxx | X |
| X | X | XX.X - XX.X | X.XXX | X |
| X | X | XX.X - XX.X | X.XXX | X |
| X | X | XX.X - XX.X | X.XXX | X |
| X | X | XX.X - XX.X | X.XXX | X |
| X | X | XX.X - XX.X | X.XXX | X |

320 mg: Administration of 320 mg (4 x 80 mg capsules) LOXO-292 on Day 1 640 mg: Administration of 640 mg (8 x 80 mg capsules) LOXO-292 on Day 1 720 mg: Administration of 720 mg (9 x 80 mg capsules) LOXO-292 on Day 1

R2 = Coefficient of determination

n = Number of points used in Kel calculation

. = Kel value not reportable.

# Notes for Generating the Actual Table:

Presentation of Data:

- Interval start and stop times will be presented to 1 decimal or 3 sig figures min;
- R2 will be presented to 3 decimals;
- n will be presented as an integer (with no decimal)

Program: /CAXXXXX/sas\_prg/pksas/kel-tables-parallel.sas DDMMYYYY HH:MM

Program: /CAXXXXX/sas\_prg/pksas/adam\_kel.sas DDMMMYYYY HH:MM

# Table 14.2.1.8 will be in the following format:

Table 14.2.1.8 Dose Proportionality Analysis of Plasma LOXO-292 Following Administration of Single Ascending Doses of LOXO-292 (Cohorts 1 - 3) (PK Population)

| Pharmacokinetic<br>Parameters | Estimate of Slope (b) | Standard<br>Error | 90% Confidence Interval<br>for Slope |
|---|---|---|---|
| Paraml | X.XXXX | X.XXXX | X.XXXX - X.XXXX |
| Param2 | X.XXXX | X.XXXX | X.XXXX - X.XXXX |
| Param3 | X.XXX | X.XXXX | X.XXXX - X.XXXX |

#### Presentation of Data:

- · Slope will be presented to 4 decimal places
- · Standard error will be presented to 4 decimal places
- 90% CI will be presented to 4 decimal places

Loxo Oncology, Inc. LOXO-292, LOXO-RET-18057 Celerion, Clinical Study Report No. CA27486

#### Notes for Generating the Actual Table:

Programmers Note:

PK Parameters are AUCO-24, AUCO-t, AUCO-inf, and Cmax

Please use the footnote below:

Parameters were ln-transformed prior to analysis.

The following statistical model using PROC MIXED of SAS was used to test dose proportionality: Parameter =  $a * Dose^b$  which was equivalent to ln(Parameter) = ln(a) + b[ln(Dose)]

Dose proportionality is not rejected if the 90% CI for b contains 1.

Program: DDMMYYYY HH:MM

Program: /CAXXXXX/sas\_prg/pksas/adam\_dosepropmixed.sas DDMMMYYYY HH:MM

Table 14.3.1.1 Treatment-emergent Adverse Event Frequency by Treatment - Number of Subjects Reporting Events (% of Subject Dosed) (Safety Population)

| TE Adverse Event* | 320 mg | 640 mg | 720 mg | Overall |
|---|---|---|---|---|
| Number of Subjects Dosed | X (100%) | X (100%) | X (100%) | X (100%) |
| Number of Subjects with TE Adverse Events | X (XX%) | X (XX%) | X (XX%) | X (XX%) |
| Number of Subjects without TE Adverse Events | X (XX%) | X (XX%) | X (XX%) | X (XX%) |
| Nervous system disorders | X (XX%) | X (XX%) | X (XX%) | X (XX%) |
| Dizziness | X (XX%) | X (XX%) | X (XX%) | X (XX%) |
| Headache | X (XX%) | X (XX%) | X (XX%) | X (XX%) |
| Presyncope | X (XX%) | X (XX%) | X (XX%) | X (XX%) |
| Respiratory, thoracic and mediastinal disorders | X (XX%) | X (XX%) | X (XX%) | X (XX%) |
| Dry throat | X (XX%) | X (XX%) | X (XX%) | X (XX%) |
| Oropharyngeal pain | X (XX%) | X (XX%) | X (XX%) | X (XX%) |
| Sinus congestion | X (XX%) | X (XX%) | X (XX%) | X (XX%) |
| Sneezing | X (XX%) | X (XX%) | X (XX%) | X (XX%) |
| etc. | | | | |

Note: \* Adverse events are classified according to MedDRA Version 21.1 by System Organ Class and Preferred Term.

TE = Treatment-emergent

For an AE with multiple changes in severity, a new record with severity less or equal to its maximum severity will not be included in the adverse event summary tables.

320 mg: Administration of 320 mg (4 x 80 mg capsules) LOXO-292 on Day 1 640 mg: Administration of 320 mg (8 x 80 mg capsules) LOXO-292 on Day 1

720 mg: Administration of 320 mg (9 x 80 mg capsules) LOXO-292 on Day 1

Program: /CAXXXXX/sas\_prg/stsas/tab\_PROGRAMNAME.sas DDMMYYYYY HH:MM

Programmer Note: Sort by decreasing frequency of system organ class and by preferred term within a system organ class of Overall column. For each subject, please sort the AEs with same verbatim and preferred term by onset date/time. For any pair (e.g., AE\_S1, AE\_S2) of these AEs (for same subject, same verbatim and preferred term), if the onset date/time of AE\_S2 = resolved date/time of AE\_S1 and the grade of AE\_S2 < the grade level of AE\_S1, then mark the AE\_S2 with a flag like EVAUL\_FLG ="N". Then, for AE analysis (summary tables), please exclude the ones with EVAUL\_FLG ="N". Won't repeat this comment again.

Page 1 of 1

Table 14.3.1.2 Treatment-Emergent Adverse Event Frequency by Treatment, Severity Grade, and Relationship to Study Drugs - Number of Subjects Reporting Events (Safety Population)

| | | Number of | S | Severi | ty Gr | ade | Relationship to Study Drug | | |
|---|---|---|---|---|---|---|---|---|---|
| TE Adverse Event* | Treatment | Subjects with<br>Adverse Events | 1 | 2 | 3 | 4 | 5 | Related | Not Related |
| Dizziness | 320 mg | X | X | X | X | X | X | X | X |
| Dry eye | 640 mg | X | X | X | X | X | X | X | X |
| Dry mouth | XXX mg | X | X | X | X | X | X | X | X |
| _ | _ | X | X | X | X | X | X | X | X |
| Dry throat | XXX mg | X | X | X | X | X | X | X | X |
| Ear pain | XXX mg | X | X | X | X | X | X | X | X |
| Fatigue | XXX mg | X | Χ | Χ | Χ | Χ | X | X | X |
| Treatment 320 mg | | XX | X | X | X | X | X | X | X |
| Treatment 640 mg | | XX | X | X | Χ | X | X | X | X |
| Treatment 720 mg | | XX | X | X | X | X | X | X | X |
| Overall | | XX | X | X | X | X | X | X | X |

Note: \* Adverse events are classified according to MedDRA Version 21.1 by System Organ Class and Preferred Term.

TE = Treatment-emergent; AE = Adverse event

Severity Grade: Grade 1 = Mild; Grade 2 = Moderate; Grade 3 = Severe or medically significant but not immediately lifethreatening; Grade 4 = Life-threatening consequences; Grade 5 = Death related to AE.

AEs are graded according to NCI CTCAE version 5.0 grading scale. Not all grades are appropriate for all AEs, therefore some AEs are listed in the CTCAE with fewer than 5 options for grade selection.

If a TEAE decreased in severity grade, the new TEAE record with less severity was counted as the same TEAE event of the previous record with worse severity under the same treatment group.

When a subject experienced the same TEAE at more than one level of severity during a treatment period, only the most severe one was counted.

When a subject experienced the same TEAE at more than one level of drug relationship during a treatment period, only the one related to study drugs was counted.

320 mg: Administration of 320 mg (4 x 80 mg capsules) LOXO-292 on Day 1  $\,$ 

640 mg: Administration of 320 mg (8 x 80 mg capsules) LOXO-292 on Day 1  $\,$ 

720 mg: Administration of 320 mg (9 x 80 mg capsules) LOXO-292 on Day 1

Table 14.3.2.1 Serious Adverse Events (Safety Population)

| Subject | | | Adverse | PT* / | Ons | et/Resoluti | on | | Severity | | | | Other<br>Action | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Number | Treatment | TE?^ | | SOC | Day | Date | Time | Freq* | Grade | Ser* | Outcome | Action | | Relationship |
| XXX-XXX | 640 mg | Yes | XXXXXXX | XXXXXXX/<br>XXXXXXXX | XX/<br>XX | DDMMYYYY/<br>DDMMYYYYY | XX:XX/<br>XX:XX | Inter. | X | NS | Recovered or resolved | XXXXXXXXXX | | XXXXXXXXX/<br>XXXXXXXXX |

Note: \* Adverse events are classified according to MedDRA Version 21.1 by System Organ Class and Preferred Term.

TE = Treatment-emergent; PT = Preferred Term; SOC = System Organ Class, Onset day is relative to Period 1 Day 1.

Freq\* represents Frequency: SI = Single Episode, Inter. = Intermittent, Cont. = Continuous

Ser\* represents Serious: NS = Not Serious

Severity/Intensity: Grade 1 = Mild; Grade 2 = Moderate; Grade 3 = Severe or medically significant but not immediately life-threatening; Grade 4 = Life-threatening consequences; Grade 5 = Death related to AE

AEs are graded according to NCI CTCAE version 5.0 grading scale. Not all grades are appropriate for all AEs, therefore some AEs are listed in the CTCAE with fewer than 5 options for grade selection.

320 mg: Administration of 320 mg (4 x 80 mg capsules) LOXO-292 on Day 1

640 mg: Administration of 320 mg (9 x 80 mg capsules) LOXO-292 on Day 1

720 mg: Administration of 320 mg (9 x 80 mg capsules) LOXO-292 on Day 1

Program: /CAXXXXX/sas prq/stsas/tab PROGRAMNAME.sas DDMMYYYYY HH:MM

Programmer Note: if there are no serious adverse events reported, there will be just one table (Table 14.3.2.1) with the statement "There was no serious adverse event recorded during the study."

# Tables 14.3.4.1-14.3.4.3 will have the following format.


| m 1 7 4 2 4 4 | 0 1 5 0 77 | 1 D 1 1 | D 11 C | C1 ' 1 | (Safety Population) |
|---|---|---|---|---|---|
| Table 14.3.4.1 | Unr-or-kange va | allies and Recheck | Kesilits - Serim | Chemistry ( | (Safety Population) |

| Subject<br>Number | Treatment | Age\$/<br>Sex | Study<br>Period | Day | Hour | Date | Parameter1<br>< Range><br>(Unit) | Parameter2<br>< Range><br>(Unit) | Parameter3<br>< Range><br>(Unit) | Parameter4<br>< Range><br>(Unit) | Parameter5<br>< Range><br>(Unit) |
|---|---|---|---|---|---|---|---|---|---|---|---|
| XXX-XXX | XXX mg | XX/M | Screen | | | DDMMYYYY | XX HN | XX | XX | XX | XX HN |
| | (Z | | 1 | -x | Check-in | DDMMYYYYY | XX | XX | XX | XX | XX |
| | | | 1 | X | X | DDMMYYYYY | XX | XX | XX | XX HN | XX |
| | | | | X | X | DDMMYYYY | XX | XX | XX | XX | XX |
| | | | | X | X | DDMMYYYY | XX LY- | XX LN | XX | XX LY- | XX |

Programmer Note: Replace Parameter1, 2 etc. with actual lab tests in the study. Sort unscheduled assessment and early term chronologically with other scheduled assessments and rechecks. Recheck should be sorted with the scheduled time point the recheck is for. Arrange alphabetically by lab test name.

Note: \$ Age is calculated from the date of first dosing

Abnormal flag: H = Above Reference Range, L = Below Reference Range

Computer Clinical significance: N = Not Clinically Significant, Y = Clinically Significant

PI Interpretation: - = Not Clinically Significant, R = To be Rechecked, ^ = Will be Retested at a Later Event

320 mg: Administration of 320 mg (4 x 80 mg capsules) LOXO-292 on Day 1

640 mg: Administration of 320 mg (8 x 80 mg capsules) LOXO-292 on Day 1

720 mg: Administration of 320 mg (9 x 80 mg capsules) LOXO-292 on Day 1

Table 14.3.4.4 Clinically Significant Laboratory and Corresponding Results (Safety Population)

| Subject<br>Number | Treatment | Age\$/<br>Sex | | Day | Hour | Date | Time | Department | Test | Result | Reference Range | Unit |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| XXX-XXX | XXX mg | XX/X | Х | Х | x.xx | DDMMYYYY | HH:MM:SS | Serum Chemistry | Cholesterol | XXX | x - x | mg/dL |
| | 0.00000000 | | | | | | | Serum Chemistry | | XXX HYR+ | X - X | mg/dL |
| | | | | | | | | Serum Chemistry | | XXX HY- | x - x | mg/dL |
| | | | | X | XX.XX | DDMMYYYYY | HH:MM:SS | Serum Chemistry | Cholesterol | XXX HN | x - x | mg/dL |

Programmer Note: All time points for a subject/test with at least one value deemed as CS by the PI will be presented in this table.

If there were no CS values as deemed by PI (i.e., no "CS" or "Clinically Significant" in the PI flag or comment field in the laboratory dataset), then this table will contain only the statement: "There were no laboratory values deemed

clinically significant by the PI in the study."

Note: \$ Age is calculated from the date of first dosing

H = Above Reference Range, L = Below Reference Range

Computer: N = Not Clinically Significant, Y = Clinically Significant

PI Interpretation: - = Not Clinically Significant, R = To be Rechecked, ^ = Will be Retested at a Later Event

320 mg: Administration of 320 mg (4 x 80 mg capsules) LOXO-292 on Day 1 640 mg: Administration of 320 mg (8 x 80 mg capsules) LOXO-292 on Day 1 720 mg: Administration of 320 mg (9 x 80 mg capsules) LOXO-292 on Day 1

# Tables 14.3.5.1, 14.3.5.3, and 14.3.5.5 will have the following format.


Table 14.3.5.1 Clinical Laboratory Summary and Change from Baseline - Serum Chemistry (Safety Population)

| | | Time | | | Treatment | 5 | Change From Bas | | |
|---|---|---|---|---|---|---|---|---|---|
| Laboratory Test (unit) | Normal Range# | | Statistic | 320 mg | 640 mg | 720 mg | | 640 mg | 720 mg |
| Parameter1 (unit) | XX - XX | Day -1 | Mean<br>SD<br>Minimum<br>Median | XX<br>XX.XX<br>X.XXX<br>XX.X<br>XX.XX<br>XX.XX | XX<br>XX.XX<br>X.XXX<br>XX.X<br>XX.X | | | | |
| | | Day 2 | n<br>Mean<br>SD<br>Minimum<br>Median<br>Maximum | XX<br>XX.XX<br>X.XXX<br>XX.X<br>XX.XX | XX<br>XX.XX<br>X.XXX<br>XX.X<br>XX.XX | XX<br>XX.XX<br>X.XXX<br>XX.X<br>XX.XX<br>XX.XX | XX<br>XX.XX<br>X.XXX<br>XX.X<br>XX.XX | XX<br>XX.XX<br>X.XXX<br>XX.X<br>XX.XX<br>XX.XX | XX<br>XX.XX<br>X.XXX<br>XX.X<br>XX.X |
| | | Day 5 | n<br>Mean<br>SD<br>Minimum<br>Median<br>Maximum | XX<br>XX.XX<br>X.XXX<br>XX.X<br>XX.XX | XX<br>XX.XX<br>X.XXX<br>XX.X<br>XX.XX | XX<br>XX.XX<br>X.XXX<br>XX.X<br>XX.X | XX<br>XX.XX<br>X.XXX<br>XX.X<br>XX.XX | XX<br>XX.XX<br>X.XXX<br>XX.XX<br>XX.XX | XX<br>XX.XX<br>X.XXX<br>XX.X<br>XX.XX |

<Programmer note: Similar for remaining laboratory tests. Also need to add Day 8 time point. Sort alphabetically by lab test name.>

Note: # Lowest of the lower ranges and highest of the higher ranges are used. Refer to Appendix 16.1.10.1 for the breakdown.

Baseline is Day -1 check-in and is the last non-missing predose measurement prior to dosing, including rechecks and unscheduled assessments.

320 mg: Administration of 320 mg (4 x 80 mg capsules) LOXO-292 on Day 1 640 mg: Administration of 320 mg (8 x 80 mg capsules) LOXO-292 on Day 1 720 mg: Administration of 320 mg (9 x 80 mg capsules) LOXO-292 on Day 1

### Tables 14.3.5.2, 14.3.5.4, and 14.3.5.6 will have the following format.


Table 14.3.5.2 Clinical Laboratory Shift from Baseline - Serum Chemistry (Safety Population)

| | | | Ва | seline | L | Bas | seline | N | Bas | eline | Н | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Laboratory | | Time - | <br>P | ostdos<br> | e<br> | <br>F | ostdo | ======<br>se<br>====== | <br>P | ostdo: | <br>se<br> | _ |
| Test (units) | Treatment | Point | L | N | Н | L | N | Н | L | N | Н | |
| Testname(unit) | XXX mg | Day 2 | Х | XX | X | Х | XX | X | Х | XX | Х | |
| | | Day 5 | Χ | XX | X | Χ | XX | X | Χ | XX | Χ | |
| | | Day 8 | Х | XX | Х | Χ | XX | Х | Χ | XX | Х | |

<Programmer note: Similar for remaining laboratory tests. Use N = Within Normal Range, O = Outside Normal Range for urinalysis shift table.>

Note: N = Within Normal Range, L = Below Normal Range, H = Above Normal Range.

Baseline is Day -1 check-in and is the last non-missing predose measurement prior to dosing of LOXO-292, including rechecks and unscheduled assessments.

320 mg: Administration of 320 mg (4 x 80 mg capsules) LOXO-292 on Day 1 640 mg: Administration of 320 mg (8 x 80 mg capsules) LOXO-292 on Day 1 720 mg: Administration of 320 mg (9 x 80 mg capsules) LOXO-292 on Day 1

Program: /CAXXXXX/sas\_prg/stsas/tab\_programname.sas DDMMMYYYY HH:MM

Table 14.3.5.7 Vital Sign Summary and Change from Baseline (Safety Population)

| **** | m.' | | 7 | Γreatment | | Change From Baseline | | |
|---|---|---|---|---|---|---|---|---|
| Vital sign<br>Paramater (unit) | Time<br>Point | Statistic | 320 mg | 640 mg | 720 mg | 320 mg | 640 mg | 720 mg |
| Parameter1 (unit) | Day -1 Check-in | Median | XX.XX<br>X.XXX<br>XX.X<br>XX.XX | XX<br>XX.XX<br>X.XXX<br>XX.X<br>XX.X | | | | |
| | Day 1 Predose | Median | XX.XX<br>X.XX<br>XX.X<br>XX.X | X.XXX<br>XX.X | | | | |
| | Day 1 Hour 2 | Mean<br>SD<br>Minimum<br>Median | X.XXX<br>XX.X<br>XX.XX | XX.XX<br>X.XXX<br>XX.X<br>XX.XX | XX.XX<br>X.XXX<br>XX.X<br>XX.X | XX<br>XX.XX<br>X.XXX<br>XX.X<br>XX.XX | XX.XX<br>X.XXX<br>XX.X | XX.XX<br>X.XXX<br>XX.X |

<Programmer note: Similar for remaining vital sign parameters. Also need to add additional time points: Day 1 Hour 4,
Day 2, Day 3, Day 4, Day 5, Day 6, Day 7, and Day 8.</pre>

Note: Baseline is Day 1 predose and is the last non-missing predose measurement prior to dosing, including rechecks and unscheduled assessments.>

320 mg: Administration of 320 mg (4 x 80 mg capsules) LOXO-292 on Day 1 640 mg: Administration of 320 mg (8 x 80 mg capsules) LOXO-292 on Day 1

720 mg: Administration of 320 mg (9 x 80 mg capsules) LOXO-292 on Day 1


Table 14.3.5.8 12-Lead Electrocardiogram Summary and Change from Baseline (Safety Population)

| | Time | | - | Γreatment | | Change From Baseline | | |
|---|---|---|---|---|---|---|---|---|
| ECG Paramater (unit) | | Statistic | 320 mg | 640 mg | 720 mg | | 640 mg | 720 mg |
| Parameter1 (unit) | Day -1 | Mean<br>SD<br>Minimum<br>Median | XX.XX<br>X.XXX<br>XX.X<br>XX.XX | | | | | |
| | Day 2 | Median | XX.XX<br>X.XXX<br>XX.X<br>XX.X | X.XXX<br>XX.X | XX.XX<br>X.XXX<br>XX.X<br>XX.XX | XX.XX<br>X.XXX<br>XX.X | X.XXX<br>XX.X | XX<br>XX.XX<br>X.XXX<br>XX.X<br>XX.X |
| | Day 5 | n<br>Mean<br>SD<br>Minimum<br>Median<br>Maximum | XX.XX<br>X.XXX<br>XX.X<br>XX.X | XX.XX<br>X.XXX<br>XX.X | | XX<br>XX.XX<br>X.XX<br>XX.X<br>XX.XX | XX<br>XX.XX<br>X.XXX<br>XX.X<br>XX.XX | XX<br>XX.XX<br>X.XXX<br>XX.X<br>XX.XX |

<Programmer note: Similar for remaining ECG parameters. Also need to add Day 8 time point.>

Note: Baseline is Day -1 check-in assessment and is the last non-missing predose measurement prior to dosing, including rechecks and unscheduled assessments.

320 mg: Administration of 320 mg (4 x 80 mg capsules) LOXO-292 on Day 1 640 mg: Administration of 320 mg (8 x 80 mg capsules) LOXO-292 on Day 1

720 mg: Administration of 320 mg (9 x 80 mg capsules) LOXO-292 on Day 1  $\,$ 

### 11. LISTING SHELLS

The following listing shells provide a framework for the display of data from this study. The shells may change due to unforeseen circumstances. These shells may not be reflective of every aspect of this study, but are intended to show the general layout of the listings that will be presented and included in the final CSR. These listings will be generated off of the Celerion SDTM Tabulation Model 1.4 mapped in accordance with SDTM Implementation Guide 3.2. All listings will be presented in Courier New size font 9.

Appendix 16.1.10.1 Clinical Laboratory Reference Ranges

| Laboratory Group | Test Name | Sex | Age Category | Normal Range | Unit |
|------------------|-----------|--------|--------------|--------------|-------|
| Serum Chemistry | Test Name | XXXXXX | XX | XX - XX | units |
| _ | Test Name | XXXXXX | XX | XX - XX | units |
| | Test Name | XXXXXX | XX | XX - XX | units |
| | Test Name | XXXXXX | XX | XX - XX | units |
| | Test Name | XXXXXX | XX | XX - XX | units |
| | Test Name | XXXXXX | XX | XX - XX | units |
| Hematology | Test Name | XXXXXX | XX | XX - XX | units |
| | Test Name | XXXXXX | XX | XX - XX | units |
| | Test Name | XXXXXX | XX | XX - XX | units |
| | Test Name | XXXXXX | XX | XX - XX | units |
| | Test Name | XXXXXX | XX | XX - XX | units |

<similar for remaining Laboratory Groups and Test Names>

<sup>&</sup>lt;Programmer note: Sort alphabetically by lab test name within each lab group.>

Appendix 16.2.1 Subject Discontinuation (Safety Population)

| Treatment | Subject<br>Number | Study<br>Period | l Date | Completed<br>Study? | Primary Discontinuation Reason |
|---|---|---|---|---|---|
| XXX mg XXX mg XXX mg XXX mg XXX mg XXX mg | XXX-XXX<br>XXX-XXX<br>XXX-XXX<br>XXX-XXX<br>XXX-XXX | Post<br>Post<br>Post<br>Post<br>Post<br>Post | DDMMYYYY<br>DDMMYYYY<br>DDMMYYYY<br>DDMMYYYY<br>DDMMYYYY<br>DDMMYYYY | YES YES YES NO YES YES | Adverse Event |

Note: 320 mg: Administration of 320 mg (4 x 80 mg capsules) LOXO-292 on Day 1 640 mg: Administration of 320 mg (8 x 80 mg capsules) LOXO-292 on Day 1 720 mg: Administration of 320 mg (9 x 80 mg capsules) LOXO-292 on Day 1

Appendix 16.2.4.1 Demographics (Safety Population)

| Treatment | Subject<br>Number | Date of<br>Birth | Age*<br>(yrs) | Sex | Race | Ethnicity | Height (cm) | Weight<br>(kg) | Body Mass<br>Index<br>(kg/m^2) | Informed<br>Consent<br>Date | Informed<br>Consent<br>Version Date |
|---|---|---|---|---|---|---|---|---|---|---|---|
| XXX mg | XXX-XXX | DDMMYYYY | XX | AAAAA | AAAAAAA | AAAAAAAAA | XXX | XX.XX | xx.xx | DDMMYYYYY | DDMMYYYY |
| XXX mg | XXX-XXX | <b>DDMMYYYYY</b> | XX | AAAAA | AAAAAAA | AAAAAAAAA | XXX | XX.XX | XX.XX | DDMMYYYYY | DDMMYYYYY |
| XXX mg | XXX-XXX | DDMMYYYY | XX | AAAAA | AAAAAAA | AAAAAAAAA | XXX | XX.XX | XX.XX | DDMMYYYYY | DDMMYYYYY |
| XXX mg | XXX-XXX | DDMMYYYY | XX | AAAAA | AAAAAAA | AAAAAAAAA | XXX | XX.XX | XX.XX | DDMMYYYYY | DDMMYYYY |
| XXX mg | XXX-XXX | <b>DDMMYYYYY</b> | XX | AAAAA | AAAAAAA | AAAAAAAAA | XXX | XX.XX | XX.XX | DDMMYYYYY | DDMMYYYY |
| XXX mg | XXX-XXX | DDMMYYYYY | XX | AAAAA | AAAAAAA | AAAAAAAA | XXX | XX.XX | XX.XX | DDMMYYYYY | DDMMYYYYY |
| XXX mg | XXX-XXX | DDMMYYYYY | XX | AAAAA | AAAAAAA | AAAAAAAA | XXX | XX.XX | XX.XX | DDMMYYYYY | DDMMYYYY |

Note: \* Age is calculated form the date of first dosing.

320 mg: Administration of 320 mg (4 x 80 mg capsules) LOXO-292 on Day 1 640 mg: Administration of 320 mg (8 x 80 mg capsules) LOXO-292 on Day 1 720 mg: Administration of 320 mg (9 x 80 mg capsules) LOXO-292 on Day 1

Appendix 16.2.4.2 Updated Informed Consent (Safety Population)

| Treatment | Subject<br>Number | Date Subject Signed<br>Informed Re-Consent | Informed Re-Consent<br>Version Date | Reason for<br>Re-Consent |
|---|---|---|---|---|
| XXX mg | XXX-XXX | DDMMYYYY | DDMMYYYYY | XXXXXXXXXXXXX |
| XXX mg | XXX-XXX | DDMMMYYYY | DDMMYYYYY | XXXXXXXXXXXXXX |
| XXX mg | XXX-XXX | DDMMMYYYY | DDMMYYYY | XXXXXXXXXXXXXX |
| XXX mg | XXX-XXX | DDMMYYYYY | DDMMYYYY | XXXXXXXXXXXXX |
| XXX mg | XXX-XXX | DDMMYYYYY | DDMMYYYY | XXXXXXXXXXXXX |
| XXX mg | XXX-XXX | DDMMYYYYY | DDMMYYYY | XXXXXXXXXXXXXXX |
| XXX mg | XXX-XXX | DDMMYYYYY | DDMMYYYY | XXXXXXXXXXXXXX |

Note: 320 mg: Administration of 320 mg (4 x 80 mg capsules) LOXO-292 on Day 1  $\,$ 

640 mg: Administration of 320 mg (8 x 80 mg capsules) LOXO-292 on Day 1

720 mg: Administration of 320 mg (9 x 80 mg capsules) LOXO-292 on Day 1

Appendix 16.2.4.3 Physical Examination (Safety Population)

| Subject<br>Number | Treatment | Period | Study<br>Day | Study<br>Hour | Date | Body<br>System | Answer or<br>Result | Comment |
|---|---|---|---|---|---|---|---|---|
| XXX-XXX | XXX mg | Screen | | | DDMMYYYY | Was PE performed?<br>General<br>HEENT<br>< > | Yes<br>Normal<br>Normal<br>< > | |
| | | 1 | -1 | Check-in | DDMMYYYY | Was PE performed?<br>HEENT<br>< > | Yes<br>Unchanged<br>< > | |

Note: 320 mg: Administration of 320 mg (4 x 80 mg capsules) LOXO-292 on Day 1

640 mg: Administration of 320 mg (8 x 80 mg capsules) LOXO-292 on Day 1  $\,$ 

720 mg: Administration of 320 mg (9 x 80 mg capsules) LOXO-292 on Day 1

# Loxo Oncology, Inc. LOXO-292, LOXO-RET-18057 Celerion, Clinical Study Report No. CA27486


Appendix 16.2.4.4 Medical and Surgical History (Safety Population)

| | | | | Date | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Treatment | Subject<br>Number H | Any<br>History? | Study<br>Period | Category | Body system | Start | End | Ongoing? | Condition or Events |
| XXX mg | XXX-XXX | XXX | Screen | Medical<br>Surgical | XXXXXXXXXX | DDMMYYYY<br>DDMMYYYY | DDMMYYYY<br>DDMMYYYYY | YES | XXXXXXX XXXXXXX XXXXXXXX |
| XXX mg | XXX-XXX | XXX | Screen | Medical | XXXXXXXXXX | DDMMYYYY | DDMMYYYY | NO | |

Note: 320 mg: Administration of 320 mg (4 x 80 mg capsules) LOXO-292 on Day 1 640 mg: Administration of 320 mg (8 x 80 mg capsules) LOXO-292 on Day 1 720 mg: Administration of 320 mg (9 x 80 mg capsules) LOXO-292 on Day 1

# Loxo Oncology, Inc. LOXO-292, LOXO-RET-18057 Celerion, Clinical Study Report No. CA27486


#### Appendix 16.2.5.1.1 Inclusion Criteria

- 1. Healthy, adult, male or female (of non-childbearing potential only), 18-55 years of age, inclusive, at screening.
- 3. <>
- 4. < >
- 5. <>

# Appendix 16.2.5.1.2 Exclusion Criteria

- 1. Is mentally of legally incapacitated or has significant emotional problems at the time of the screening visit or expected during the conduct of the study.

  2. <>
- 3. <>
- 4. <>
- 5. <> 6. <>
- 7. <>


# Appendix 16.2.5.2 Subject Eligibility (Safety Population)

| Treatment | Subject<br>Number | Study<br>Period | Did subject meet all eligibility criteria? | Specify |
|---|---|---|---|---|
| XXX mg | XXX-XXX | Screen | YES | |
| XXX mg | XXX-XXX | Screen | NO | <pre><this column="" data="" if="" is="" only="" present="" presented=""></this></pre> |

Note: 320 mg: Administration of 320 mg (4 x 80 mg capsules) LOXO-292 on Day 1 640 mg: Administration of 320 mg (8 x 80 mg capsules) LOXO-292 on Day 1 720 mg: Administration of 320 mg (9 x 80 mg capsules) LOXO-292 on Day 1

Page 1 of 1

Appendix 16.2.5.3.1 Check-in Criteria

1. Did the Subject report any study restriction violations since the last study visit?


# Appendix 16.2.5.3.2 Check-in Responses (Safety Population)

| Treatment | Subject<br>Number | Study<br>Period Day | Hour | Date | Time | Check-in Criteria | Specify |
|---|---|---|---|---|---|---|---|
| XXX mg | XXX-XXX | 1 X | Check-in | DDMMYYYY | hh:mm | YES | <pre><this column="" data="" if="" is="" only="" present="" prints=""></this></pre> |

Note: 320 mg: Administration of 320 mg (4 x 80 mg capsules) LOXO-292 on Day 1 640 mg: Administration of 320 mg (8 x 80 mg capsules) LOXO-292 on Day 1 720 mg: Administration of 320 mg (9 x 80 mg capsules) LOXO-292 on Day 1


# Appendix 16.2.5.4.1 Test Compound Description

| Compound | Form | Route |
|--------------|------|-------|
| XXXXXXXXXXX | < > | XXXX |
| XXXXXXXXXXXX | < > | XXXX |


# Appendix 16.2.5.4.2 Test Compound Administration Times (Safety Population)

| Treatment | Subject<br>Number | - | Day | Hour | Start<br>Date | Start<br>Time | Compound | Dosage | Comments |
|---|---|---|---|---|---|---|---|---|---|
| XXX mg | XXX-XXX | 1 | X | 0 | DDMMYYYY | HH:MM:SS | XXXXXXXX | < > | <pre><only are<br="" if="" populate="" there="">comments present in the data&gt;</only></pre> |

Note: 320 mg: Administration of 320 mg (4 x 80 mg capsules) LOXO-292 on Day 1 640 mg: Administration of 320 mg (8 x 80 mg capsules) LOXO-292 on Day 1 720 mg: Administration of 320 mg (9 x 80 mg capsules) LOXO-292 on Day 1


Appendix 16.2.5.5 PK Blood Draw Times (Safety Population)

| Subject<br>Number | Treatment | Study<br>Period | Day | Hour | Date | Actual<br>Time | Bioassay | Comments |
|---|---|---|---|---|---|---|---|---|
| XXX-XXX | XXX mg | 1 | 1 | -X.XX | DDMMYYYY | X:XX:XX | XXXXXXXXXXX | |
| | <u></u> | | | XX.XX | DDMMYYYYY | X:XX:XX | XXXXXXXXXX | |
| | | | | XX.XX | DDMMMYYYY | X:XX:XX | XXXXXXXXXX | |
| | | | | XX.XX | DDMMMYYYY | XX:XX:XX | XXXXXXXXXX | |
| | | | | XX.XX | DDMMMYYYY | XX:XX:XX | XXXXXXXXXX | |
| | | | | XX.XX | DDMMYYYYY | XX:XX:XX | XXXXXXXXXX | |
| | | | | XX.XX | DDMMMYYYY | XX:XX:XX | XXXXXXXXXX | |
| | | | | XX.XX | DDMMYYYYY | XX:XX:XX | XXXXXXXXXX | |
| | | | | XX.XX | DDMMMYYYY | XX:XX:XX | XXXXXXXXXX | |
| | | | 2 | XX.XX | DDMMMYYYY | X:XX:XX | XXXXXXXXXX | |
| | | | | XX.XX | DDMMYYYYY | X:XX:XX | XXXXXXXXXX | |
| | | | | XX.XX | DDMMYYYYY | XX:XX:XX | XXXXXXXXXX | |
| | | | 3 | XX.XX | DDMMMYYYY | X:XX:XX | XXXXXXXXXX | |

Note: 320 mg: Administration of 320 mg (4 x 80 mg capsules) LOXO-292 on Day 1

640 mg: Administration of 320 mg (8 x 80 mg capsules) LOXO-292 on Day 1

720 mg: Administration of 320 mg (9 x 80 mg capsules) LOXO-292 on Day 1


Appendix 16.2.5.6 Meal Times (Safety Population)

| Subject<br>Number | Treatment | Study<br>Period | Day | Hour | Event | Date | Start<br>Time | Stop<br>Time | Comments |
|---|---|---|---|---|---|---|---|---|---|
| XXX-XXX | XXX mg | 1 | -X<br>X<br>X | -XX.XX<br>-XX.XX<br>XX.XX<br>-XX.XX<br>XX.XX<br>-XX.XX | LUNCH<br>DINNER<br>SNACK<br>BREAKFAST | DDMMYYYY | XX:XX:XX<br>XX:XX:XX<br>XX:XX:XX<br>XX:XX:XX<br>XX:XX:XX | XX:XX:XX<br>XX:XX:XX<br>XX:XX:XX<br>XX:XX:XX<br>XX:XX: | |

Note: 320 mg: Administration of 320 mg (4 x 80 mg capsules) LOXO-292 on Day 1 640 mg: Administration of 320 mg (8 x 80 mg capsules) LOXO-292 on Day 1 720 mg: Administration of 320 mg (9 x 80 mg capsules) LOXO-292 on Day 1


# Appendix 16.2.5.7 Prior and Concomitant Medications (Safety Population)

| Subject<br>Number | Treat-<br>ment | 4 | Medication<br>(WHO* Term) | Dosage | Route | Frequency | Start<br>Day/Date/Time | Stop<br>Day/Date/Time | | • | Continuing Medication? |
|---|---|---|---|---|---|---|---|---|---|---|---|
| XXX-XXX<br>XXX-XXX | X<br>X | No<br>Yes | None<br>ACETAMINOPHEN<br>(ACETAMINOPHEN | | BY MOUTH | AS NEEDED | XX/DDMMMYYYY/<br>HH:MM | XX/DDMMYYYY/<br>HH:MM | XXXXX | XXX | YES |

Note: \* Concomitant medications are coded with WHO Dictionary Version 01SEP2018.

^ Med = Medication; UNK = Unknown

Prior medication was medication taken prior to study drug administration.

Start and stop day is relative to Period 1 Day 1.

320 mg: Administration of 320 mg (4  $\times$  80 mg capsules) LOXO-292 on Day 1

640 mg: Administration of 320 mg (8 x 80 mg capsules) LOXO-292 on Day 1

720 mg: Administration of 320 mg (9  $\times$  80 mg capsules) LOXO-292 on Day 1


# Appendix 16.2.7.1 Adverse Events (I of II) (Safety Population)

| Culadaat | | | Adriana Errent / | Time from<br>Last Dose | | Onset | | | Resolved | | Duration |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject<br>Number | Treatment | TE?^ | Adverse Event/<br>Preferred Term* | (DD:HH:MM) | Day | Date | Time | Day | Date | Time | (DD:HH:MM) |
| XXX-XXX | XXX mg | None | | | | | | | | | |
| XXX-XXX | XXX mg | Yes | XXXXXXXXXXXX/<br>XXXXXXXXXX | XX:XX:XX | XX | DDMMYYYY | X:XX | XX | DDMMYYYY | X:XX | XX:XX:XX |
| | | No | XXXXXXXXXXXXX/<br>XXXXXXXXXX | XX:XX:XX | XX | DDMMYYYY | X:XX | XX | DDMMYYYY | X:XX | XX:XX:XX |

Note: \* Adverse events are classified according to MedDRA Version 21.1 by System Organ Class and Preferred Term.

<sup>^</sup> TE = Treatment-emergent, Onset and resolved day is relative to Period 1 Day 1.

<sup>320</sup> mg: Administration of 320 mg (4 x 80 mg capsules) LOXO-292 on Day 1  $\,$ 

<sup>640</sup> mg: Administration of 320 mg (8 x 80 mg capsules) LOXO-292 on Day 1  $\,$ 

<sup>720</sup> mg: Administration of 320 mg (9 x 80 mg capsules) LOXO-292 on Day 1  $\,$ 


# Appendix 16.2.7.2 Adverse Events (II of II) (Safety Population)

| Subject | | Adverse | | Onset | | | | | | | Other<br>Action | Relationship to |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Number | Treatment | Event | Day | Date | Time | Freq* | Severity | Ser* | Outcome | Action | Taken | Study Drug |
| XXX-XXX | XXX mg | None | | | | | | | | | | |
| XXX-XXX | XXX mg | XXXXXXX | XX | DDMMYYYY | XX:XX | Inter. | Grade 1 | NO | Resolved | Dose Not<br>Changed | None | |

Note: Ser\* = Serious; Freq\* represents Frequency: SI = Single Episode, Inter. = Intermittent, Cont. = Continuous Severity/Intensity: Grade 1 = Mild; Grade 2 = Moderate; Grade 3 = Severe or medically significant but not immediately life-threatening; Grade 4 = Life-threatening consequences; Grade 5 = Death related to AE

AEs are graded according to NCI CTCAE version 5.0 grading scale. Not all grades are appropriate for all AEs, therefore some AEs are listed in the CTCAE with fewer than 5 options for grade selection.

320 mg: Administration of 320 mg (4 x 80 mg capsules) LOXO-292 on Day 1

640 mg: Administration of 320 mg (8 x 80 mg capsules) LOXO-292 on Day 1

720 mg: Administration of 320 mg (9 x 80 mg capsules) LOXO-292 on Day 1


Appendix 16.2.7.3 Adverse Event Non-Drug Therapy (Safety Population)

| 0.1.1 | | 70 -1 | | Onset | | | Resolved | | Therapy | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject<br>Number | Treatment | Adverse<br>Event | Day | Date | Time | Day | Date | Time | Date | Time | Description |
| XXX-XXX | XXX ma | DRY LIPS | XX | DDMMYYYY | X:XX | XX | DDMMYYYY | X:XX | DDMMYYYY | XX:XX | PETROLEUM JELLY |

Note: Onset and resolved day is relative to Period 1 Day 1.

320 mg: Administration of 320 mg (4 x 80 mg capsules) LOXO-292 on Day 1 640 mg: Administration of 320 mg (8 x 80 mg capsules) LOXO-292 on Day 1 720 mg: Administration of 320 mg (9 x 80 mg capsules) LOXO-292 on Day 1


# Appendix 16.2.7.4 Adverse Event Preferred Term Classification (Safety Population)

| | | | | | | Oriset | |
|---|---|---|---|---|---|---|---|
| Subject | | Adverse | | | | | |
| Number | Treatment | Event | Preferred Term* | Body System | Day | Date | Time |
| XXX-XXX | XXX mg | XXXXXX XXXXX XXXX XXXXX | XXXXXXXXXX XXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XX | DDMMYYYYY | X:XX |

Note: \* Adverse events are classified to MedDRA Version 21.1 by System Organ Class and Preferred Term.
Onset day is relative to Period 1 Day 1.

320 mg: Administration of 320 mg (4 x 80 mg capsules) LOXO-292 on Day 1 640 mg: Administration of 320 mg (8 x 80 mg capsules) LOXO-292 on Day 1 720 mg: Administration of 320 mg (9 x 80 mg capsules) LOXO-292 on Day 1

# Appendices 16.2.8.1.2-16.2.8.1.5 will have the following format.


# Appendix 16.2.8.1.1 Clinical Laboratory Report - Serum Chemistry (Safety Population)

| Cohort | Subject<br>Number | Age\$/<br>Sex | Study<br>Period | Day | Hour | Date | Parameter1<br>< Range><br>(Unit) | Parameter2<br>< Range><br>(Unit) | Parameter3<br>< Range><br>(Unit) | Parameter4<br>< Range><br>(Unit) | Parameter5<br>< Range><br>(Unit) |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Х | XXX-XXX | XX/M | Screen | | | DDMMYYYYY | XX HN | XX | XX | XX | XX HN |
| | | | 1 | -X | Check-in | <b>DDMMYYYY</b> | XX | XX | XX | XX | XX |
| | | | | X | 0 | DDMMYYYY | XX | XX | XX | XX HN | XX |
| | | | | X | 0 | DDMMYYYYY | XX | XX | XX | XX | XX |
| | | | | X | 0 | DDMMYYYY | XX LY- | XX LN | XX | XX LY- | XX |

Programmer Note: Replace Parameter1, 2 etc. with actual lab tests in the study. Sort unscheduled assessment and early term chronologically with other scheduled assessments and rechecks. Recheck should be sorted with the scheduled time point the recheck is for. Arrange alphabetically by lab test name.

Note: \$ Age is calculated from the date of first dosing.

H = Above Reference Range, L = Below Reference Range

Computer Clinical Significance: N = Not Clinically Significant, Y = Clinically Significant

PI Interpretation: - = Not Clinically Significant, R = To be Rechecked, ^ = Will be Retested at a Later Event

320 mg: Administration of 320 mg (4 x 80 mg capsules) LOXO-292 on Day 1  $\,$ 

640 mg: Administration of 320 mg (8 x 80 mg capsules) LOXO-292 on Day 1

720 mg: Administration of 320 mg (9 x 80 mg capsules) LOXO-292 on Day 1


# Appendix 16.2.8.1.6 Clinical Laboratory Report - Comments (Safety Population)

| Subject<br>Number | Treatment | Study<br>Period | Day | Hour | Date | Department | Test | Result | Unit | Comment |
|---|---|---|---|---|---|---|---|---|---|---|
| XXX-XXX | XXX mg | X | Х | -X.X | DDMMYYYY | Other Tests | Fibrinogen | XXX | mg/dL | Not significant in the context of this study. |

Note: 320 mg: Administration of 320 mg (4 x 80 mg capsules) LOXO-292 on Day 1 640 mg: Administration of 320 mg (8 x 80 mg capsules) LOXO-292 on Day 1 720 mg: Administration of 320 mg (9 x 80 mg capsules) LOXO-292 on Day 1


Appendix 16.2.8.2 Vital Signs (Safety Population)

| | | | | | | Blood 1 | Pres | sure (mmHg) | Heart | Temper- | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject<br>Number | Treat-<br>ment | Study<br>Period Day | Hour | Date | Time | | | Sys/Dia | rate<br>(bpm) | ature<br>(°C) | Weight<br>(kg) | Comments |
| XXX-XXX | XXX mg | Screen | | DDMMYYYY | X:XX:XX | | | | | | XXX.X | |
| | _ | | | DDMMYYYYY | X:XX:XX | SUPX Ri | ght | XXX/ XX | XX | XX.X | | |
| | | 1 -X | Check-in | DDMMYYYYY | XX:XX:XX | | | | | | XXX.X | |
| | | | | DDMMYYYYY | XX:XX:XX | SUPX Ri | ght | XXX/ XX | XX | | | |
| | | X | X.X | DD <b>MM</b> YYYYY | XX:XX:XX | SUPX Ri | ght | | | | | |
| | | | X.X | DD <b>MM</b> YYYYY | XX:XX:XX | SUPX Ri | ght | | | | | |
| | | | X.X | DD <b>MM</b> YYYYY | X:XX:XX | SUPX Ri | ght | XXX/ XX | XX | | | |
| | | | X.X | DD <b>MM</b> YYYYY | X:XX:XX | SUPX Ri | ght | XXX/ XX | XX | | | |
| | | | X.X | DD <b>MM</b> YYYYY | X:XX:XX | SUPX Ri | ght | XXX/ XX | XX | | | |
| | | | R | DDMMYYYYY | XX:XX:XX | SUPX Ri | ght | XXX/ XX | XX | | | |
| | | | X.X | DDMMYYYYY | XX:XX:XX | SUPX Ric | ght | | | | | |

Programmer note: Sort unscheduled assessment and early term chronologically with other scheduled assessments and rechecks. Recheck should be sorted with the scheduled time point the recheck is for.

Note: SUPX = X-minute supine, R = Recheck Value, Sys/Dia = Systolic/Diastolic 320 mg: Administration of 320 mg (4 x 80 mg capsules) LOXO-292 on Day 1 640 mg: Administration of 320 mg (8 x 80 mg capsules) LOXO-292 on Day 1 720 mg: Administration of 320 mg (9 x 80 mg capsules) LOXO-292 on Day 1


Appendix 16.2.8.3 12-Lead Electrocardiogram (Safety Population)

| Subject<br>Number | Treatment | Study<br>Period | Day | Hour | Date | Time | Result | Heart<br>Rate<br>(bpm) | PR<br>(msec) | QRS<br>(msec) | QT<br>(msec) | QTcF*<br>(msec) | Comments |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| XXX-XXX | XXX mg | Screen | | | DDMMYYYY | X:XX:XX | NORMAL | XX | XXX.X | XX.X | XXX.X | XXX.X | |
| | The state of the s | 1 | -1 | Check-in | DDMMYYYYY | X:XX:XX | NORMAL | XX | XXX.X | XX.X | XXX.X | XXX.X | |
| | | | | X.XX | <b>DDMMYYYYY</b> | X:XX:XX | NORMAL | XX | XXX.X | XX.X | XXX.X | XXX.X | |
| | | | X | X.XX | DDMMYYYYY | X:XX:XX | NORMAL | XX | XXX.X | XX.X | XXX.X | XXX.X | |
| | | | | X.XX | DDMMMYYYY | X:XX:XX | NORMAL | XX | XXX.X | XX.X | XXX.X | XXX.X | |
| | | | X | X.XX | DDMMMYYYYY | X:XX:XX | NORMAL | XX | XXX.X | XX.X | XXX.X | XXX.X # | |
| | | | X | X.XX | DDMMYYYYY | X:XX:XX | NORMAL | XX | XXX.X | XX.X | XXX.X | XXX.X @ | |

Programmer note: Sort unscheduled assessment and early term chronologically with other scheduled assessments and rechecks. Recheck should be sorted with the scheduled time point the recheck is for.

```
Note: NCS = Abnormal, Not Clinically Significant
QTcF* = QT corrected for heart rate using Fridericia's correction.
# = QTcF > 450, @ = QTcF change from baseline greater than 30 msec
320 mg: Administration of 320 mg (4 x 80 mg capsules) LOXO-292 on Day 1
640 mg: Administration of 320 mg (8 x 80 mg capsules) LOXO-292 on Day 1
720 mg: Administration of 320 mg (9 x 80 mg capsules) LOXO-292 on Day 1
```


# Appendix 16.2.8.4 Phone Call (Safety Population)

| Subject<br>Number | Treatment | Study<br>Period | Day | Phone Call Completed? | Date | Time | If no, reason |
|---|---|---|---|---|---|---|---|
| XXX-XXX | XXX ma | X | X | Yes/No | DDMMYYYYY | HH:MM | Wrong number |

Note: 320 mg: Administration of 320 mg (4 x 80 mg capsules) LOXO-292 on Day 1 640 mg: Administration of 320 mg (8 x 80 mg capsules) LOXO-292 on Day 1 720 mg: Administration of 320 mg (9 x 80 mg capsules) LOXO-292 on Day 1

# 16.1.9.2 Statistical Outputs

# Dose Proportionality Analysis for Plasma LOXO-292 PK Parameter AUCO-24 for Table 14.2.1.8 (Quadratic)

# The Mixed Procedure

#### Model Information

Data Set WORK.TOTAL
Dependent Variable LAUC24
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method
Fixed Effects SE Method
Degrees of Freedom Method Residual

### Dimensions

| Covariance Parameters | 1 |
|-----------------------|----|
| Columns in X | 3 |
| Columns in Z | 0 |
| Subjects | 1 |
| Max Obs Per Subject | 18 |

### Number of Observations

| Number | of | Observations | Read | 18 |
|--------|----|--------------|-----------|----|
| Number | of | Observations | Used | 18 |
| Number | of | Observations | Not. Used | 0 |

# Covariance Parameter Estimates

Cov Parm Estimate

Residual 0.3375

# Dose Proportionality Analysis for Plasma LOXO-292 PK Parameter AUCO-24 for Table 14.2.1.8 (Quadratic)

# The Mixed Procedure

### Fit Statistics

| -2 Res Log Likelihood | 26.2 |
|--------------------------|------|
| AIC (smaller is better) | 28.2 |
| AICC (smaller is better) | 28.5 |
| BIC (smaller is better) | 28.9 |

# Type 1 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|-------------|-----------|-----------|---------|--------|
| LDOSE | 1 | 15 | 2.60 | 0.1279 |
| LDOSE*LDOSE | 1 | 15 | 0.09 | 0.7681 |

# Dose Proportionality Analysis for Plasma LOXO-292 - AUCO-24 for Table 14.2.1.8 (Linear)

# The Mixed Procedure

#### Model Information

Data Set WORK.TOTAL
Dependent Variable LAUC24
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method
Fixed Effects SE Method
Degrees of Freedom Method Residual

### Dimensions

| Covariance Parameters | 1 |
|-----------------------|----|
| Columns in X | 2 |
| Columns in Z | 0 |
| Subjects | 1 |
| Max Obs Per Subject | 18 |

### Number of Observations

| Number | of | Observations | Read | 18 |
|--------|----|--------------|-----------|----|
| Number | of | Observations | Used | 18 |
| Number | of | Observations | Not. Used | 0 |

Covariance Parameter Estimates

Cov Parm Estimate

Residual 0.3183

# Dose Proportionality Analysis for Plasma LOXO-292 - AUCO-24 for Table 14.2.1.8 (Linear)

# The Mixed Procedure

### Fit Statistics

| -2 Res Log Likelihood | 30.8 |
|--------------------------|------|
| AIC (smaller is better) | 32.8 |
| AICC (smaller is better) | 33.1 |
| BIC (smaller is better) | 33.6 |

# Solution for Fixed Effects

| Effect | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
|---|---|---|---|---|---|---|---|---|
| Intercept | 6.3992 | 2.3343 | 16 | 2.74 | 0.0145 | 0.1 | 2.3238 | 10.4746 |
| LDOSE | 0.6169 | 0.3717 | 16 | 1.66 | 0.1165 | 0.1 | -0.03208 | 1.2658 |

# Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|--------|-----------|-----------|---------|--------|
| LDOSE | 1 | 16 | 2.75 | 0.1165 |


# Dose Proportionality Analysis for Plasma LOXO-292 - AUCO-24 for Table 14.2.1.8 (Linear)

| Parameter | Estimate | Lower<br>Limit | Upper<br>Limit |
|-----------|----------|----------------|----------------|
| Intercept | 6.3992 | 2.3238 | 10.4746 |
| Slope | 0.6169 | -0.03208 | 1.2658 |

# Dose Proportionality Analysis for Plasma LOXO-292 PK Parameter AUCO-t for Table 14.2.1.8 (Quadratic)

# The Mixed Procedure

#### Model Information

Data Set WORK.TOTAL
Dependent Variable LAUCLST
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method
Fixed Effects SE Method
Degrees of Freedom Method Residual

### Dimensions

| Covariance Parameters | 1 |
|-----------------------|----|
| Columns in X | 3 |
| Columns in Z | 0 |
| Subjects | 1 |
| Max Obs Per Subject | 18 |

### Number of Observations

| Number | of | Observations | Read | 18 |
|--------|----|--------------|-----------|----|
| Number | of | Observations | Used | 18 |
| Number | of | Observations | Not. Used | 0 |

# Covariance Parameter Estimates

Cov Parm Estimate

Residual 0.2431

# Dose Proportionality Analysis for Plasma LOXO-292 PK Parameter AUCO-t for Table 14.2.1.8 (Quadratic)

# The Mixed Procedure

### Fit Statistics

| -2 Res Log Likelihood | 21.3 |
|--------------------------|------|
| AIC (smaller is better) | 23.3 |
| AICC (smaller is better) | 23.6 |
| BIC (smaller is better) | 24.0 |

# Type 1 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|-------------|-----------|-----------|---------|--------|
| LDOSE | 1 | 15 | 3.38 | 0.0859 |
| LDOSE*LDOSE | 1 | 15 | 0.18 | 0.6797 |

# Dose Proportionality Analysis for Plasma LOXO-292 - AUCO-t for Table 14.2.1.8 (Linear)

# The Mixed Procedure

#### Model Information

Data Set WORK.TOTAL
Dependent Variable LAUCLST
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method
Fixed Effects SE Method
Degrees of Freedom Method Residual

### Dimensions

| Covariance Parameters | 1 |
|-----------------------|----|
| Columns in X | 2 |
| Columns in Z | 0 |
| Subjects | 1 |
| Max Obs Per Subject | 18 |

### Number of Observations

| Number | of | Observations | Read | 18 |
|--------|----|--------------|----------|----|
| Number | of | Observations | Used | 18 |
| Number | of | Observations | Not Used | 0 |

# Covariance Parameter Estimates

Cov Parm Estimate

Residual 0.2306

# Dose Proportionality Analysis for Plasma LOXO-292 - AUCO-t for Table 14.2.1.8 (Linear)

# The Mixed Procedure

### Fit Statistics

| -2 Res Log Likelihood | 25.7 |
|--------------------------|------|
| AIC (smaller is better) | 27.7 |
| AICC (smaller is better) | 27.9 |
| BIC (smaller is better) | 28.4 |

# Solution for Fixed Effects

| Effect | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
|---|---|---|---|---|---|---|---|---|
| Intercept | 7.0351 | 1.9866 | 16 | 3.54 | 0.0027 | 0.1 | 3.5667 | 10.5035 |
| LDOSE | 0.5970 | 0.3163 | 16 | 1.89 | 0.0774 | 0.1 | 0.04475 | 1.1493 |

# Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|--------|-----------|-----------|---------|--------|
| LDOSE | 1 | 16 | 3.56 | 0.0774 |


# Dose Proportionality Analysis for Plasma IOXO-292 - AUCO-t for Table 14.2.1.8 (Linear)

| Parameter | Estimate | Lower<br>Limit | Upper<br>Limit |
|-----------|----------|----------------|----------------|
| Intercept | 7.0351 | 3.5667 | 10.5035 |
| Slope | 0.5970 | 0.04475 | 1.1493 |

# Dose Proportionality Analysis for Plasma LOXO-292 PK Parameter AUCO-inf for Table 14.2.1.8 (Quadratic)

# The Mixed Procedure

#### Model Information

Data Set WORK.TOTAL
Dependent Variable LAUCIFO
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method
Fixed Effects SE Method
Degrees of Freedom Method Residual

### Dimensions

| Covariance Parameters | 1 |
|-----------------------|----|
| Columns in X | 3 |
| Columns in Z | 0 |
| Subjects | 1 |
| Max Obs Per Subject | 18 |

### Number of Observations

| Number | of | Observations | Read | 18 |
|--------|----|--------------|-----------|----|
| Number | of | Observations | Used | 18 |
| Number | of | Observations | Not. Used | 0 |

# Covariance Parameter Estimates

Cov Parm Estimate

Residual 0.2437

# Dose Proportionality Analysis for Plasma LOXO-292 PK Parameter AUCO-inf for Table 14.2.1.8 (Quadratic)

# The Mixed Procedure

### Fit Statistics

| -2 Res Log Likelihood | 21.3 |
|--------------------------|------|
| AIC (smaller is better) | 23.3 |
| AICC (smaller is better) | 23.6 |
| BIC (smaller is better) | 24.0 |

# Type 1 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|-------------|-----------|-----------|---------|--------|
| LDOSE | 1 | 15 | 3.39 | 0.0854 |
| LDOSE*LDOSE | 1 | 15 | 0.18 | 0.6790 |

# Dose Proportionality Analysis for Plasma LOXO-292 - AUCO-inf for Table 14.2.1.8 (Linear)

# The Mixed Procedure

#### Model Information

Data Set WORK.TOTAL
Dependent Variable LAUCIFO
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method
Fixed Effects SE Method
Degrees of Freedom Method Residual

### Dimensions

| Covariance Parameters | 1 |
|-----------------------|----|
| Columns in X | 2 |
| Columns in Z | 0 |
| Subjects | 1 |
| Max Obs Per Subject | 18 |

### Number of Observations

| Number | of | Observations | Read | 18 |
|--------|----|--------------|-----------|----|
| Number | of | Observations | Used | 18 |
| Number | of | Observations | Not. Used | 0 |

# Covariance Parameter Estimates

Cov Parm Estimate

Residual 0.2312

# Dose Proportionality Analysis for Plasma LOXO-292 - AUCO-inf for Table 14.2.1.8 (Linear)

# The Mixed Procedure

### Fit Statistics

| -2 Res Log Likelihood | 25.7 |
|--------------------------|------|
| AIC (smaller is better) | 27.7 |
| AICC (smaller is better) | 28.0 |
| BIC (smaller is better) | 28.5 |

# Solution for Fixed Effects

| Effect | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
|---|---|---|---|---|---|---|---|---|
| Intercept | 7.0292 | 1.9893 | 16 | 3.53 | 0.0028 | 0.1 | 3.5561 | 10.5023 |
| LDOSE | 0.5990 | 0.3168 | 16 | 1.89 | 0.0769 | 0.1 | 0.04592 | 1.1520 |

# Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|--------|-----------|-----------|---------|--------|
| LDOSE | 1 | 16 | 3.58 | 0.0769 |


# Dose Proportionality Analysis for Plasma LOXO-292 - AUCO-inf for Table 14.2.1.8 (Linear)

| Parameter | Estimate | Lower<br>Limit | Upper<br>Limit |
|-----------|----------|----------------|----------------|
| Intercept | 7.0292 | 3.5561 | 10.5023 |
| Slope | 0.5990 | 0.04592 | 1.1520 |

# Dose Proportionality Analysis for Plasma LOXO-292 PK Parameter Cmax for Table 14.2.1.8 (Quadratic)

# The Mixed Procedure

#### Model Information

Data Set WORK.TOTAL
Dependent Variable LCMAX
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method
Fixed Effects SE Method
Degrees of Freedom Method Residual

### Dimensions

| Covariance Parameters | 1 |
|-----------------------|----|
| Columns in X | 3 |
| Columns in Z | 0 |
| Subjects | 1 |
| Max Obs Per Subject | 18 |

### Number of Observations

| Number | of | Observations | Read | 18 |
|--------|----|--------------|-----------|----|
| Number | of | Observations | Used | 18 |
| Number | of | Observations | Not. Used | 0 |

# Covariance Parameter Estimates

Cov Parm Estimate

Residual 0.3736

# Dose Proportionality Analysis for Plasma LOXO-292 PK Parameter Cmax for Table 14.2.1.8 (Quadratic)

# The Mixed Procedure

### Fit Statistics

| -2 Res Log Likelihood | 27.7 |
|--------------------------|------|
| AIC (smaller is better) | 29.7 |
| AICC (smaller is better) | 30.1 |
| BIC (smaller is better) | 30.5 |

# Type 1 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|-------------|-----------|-----------|---------|--------|
| LDOSE | 1 | 15 | 2.12 | 0.1662 |
| LDOSE*LDOSE | 1 | 15 | 0.02 | 0.8827 |
## Dose Proportionality Analysis for Plasma LOXO-292 - Cmax for Table 14.2.1.8 (Linear)

#### The Mixed Procedure

#### Model Information

Data Set WORK.TOTAL
Dependent Variable LCMAX
Covariance Structure Diagonal
Estimation Method REML
Residual Variance Method
Fixed Effects SE Method
Degrees of Freedom Method Residual

#### Dimensions

| Covariance Parameters | 1 |
|-----------------------|----|
| Columns in X | 2 |
| Columns in Z | 0 |
| Subjects | 1 |
| Max Obs Per Subject | 18 |

#### Number of Observations

| Number | of | Observations | Read | 18 |
|--------|----|--------------|-----------|----|
| Number | of | Observations | Used | 18 |
| Number | of | Observations | Not. Used | 0 |

### Covariance Parameter Estimates

Cov Parm Estimate

Residual 0.3508

## Dose Proportionality Analysis for Plasma LOXO-292 - Cmax for Table 14.2.1.8 (Linear)

#### The Mixed Procedure

#### Fit Statistics

| -2 Res Log Likelihood | 32.4 |
|--------------------------|------|
| AIC (smaller is better) | 34.4 |
| AICC (smaller is better) | 34.7 |
| BIC (smaller is better) | 35.1 |

#### Solution for Fixed Effects

| Effect | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
|---|---|---|---|---|---|---|---|---|
| Intercept | 4.3482 | 2.4504 | 16 | 1.77 | 0.0950 | 0.1 | 0.07012 | 8.6262 |
| LDOSE | 0.5860 | 0.3902 | 16 | 1.50 | 0.1526 | 0.1 | -0.09519 | 1.2673 |

#### Type 3 Tests of Fixed Effects

| Effect | Num Den<br>DF DF | | F Value | Pr > F |
|--------|------------------|----|---------|--------|
| LDOSE | 1 | 16 | 2.26 | 0.1526 |


# Dose Proportionality Analysis for Plasma LOXO-292 - Cmax for Table 14.2.1.8 (Linear)

| Parameter | Estimate | Lower<br>Limit | Upper<br>Limit |
|-----------|----------|----------------|----------------|
| Intercept | 4.3482 | 0.07012 | 8.6262 |
| Slope | 0.5860 | -0.09519 | 1.2673 |

# Dose Proportionality Analysis for Plasma LOXO-292 - AUCO-t for Figure 14.2.2.7

Model: MODEL1

Dependent Variable: AVAL Analysis Value

Number of Observations Read 18 Number of Observations Used 18

#### Analysis of Variance

| Source | | DF | Sum of<br>Squares | Mean<br>Square | F Value | Pr > F |
|---|---|---|---|---|---|---|
| Model<br>Error<br>Corrected Total | | 1<br>16<br>17 | 0.82125<br>3.68893<br>4.51018 | 0.82125<br>0.23056 | 3.56 | 0.0774 |
| | Root MSE<br>Dependent M<br>Coeff Var | ean | 0.48016<br>10.77842<br>4.45487 | R-Square<br>Adj R-Sq | 0.1821<br>0.1310 | |

# Dose Proportionality Analysis for Plasma LOXO-292 - AUCO-t for Figure 14.2.2.7

Model: MODEL1

Dependent Variable: AVAL Analysis Value

Parameter Estimates

| Variable | Label | DF | Parameter<br>Estimate | Standard<br>Error | t Value | Pr > t |
|---|---|---|---|---|---|---|
| Intercept | Intercept Log Value of Actual Treatment | 1 | 7.03512 | 1.98661 | 3.54 | 0.0027 |
| LDOSE | | 1 | 0.59705 | 0.31635 | 1.89 | 0.0774 |

# Dose Proportionality Analysis for Plasma LOXO-292 - AUCO-t for Figure 14.2.2.7

Model: MODEL1 Dependent Variable: AVAL Analysis Value

#### Output Statistics

| Obs | Dependent<br>Variable | Predicted<br>Value | Std Error<br>Mean Predict | 90% CL P | redict | Residual |
|---|---|---|---|---|---|---|
| 1 | 10.4651 | 10.4791 | 0.1948 | 9.5744 | 11.3838 | -0.0140 |
| 2 | 11.1581 | 10.4791 | 0.1948 | 9.5744 | 11.3838 | 0.6791 |
| 3 | 10.9136 | 10.4791 | 0.1948 | 9.5744 | 11.3838 | 0.4345 |
| 4 | 9.5716 | 10.4791 | 0.1948 | 9.5744 | 11.3838 | -0.9075 |
| 5 | 10.2653 | 10.4791 | 0.1948 | 9.5744 | 11.3838 | -0.2138 |
| 6 | 10.5566 | 10.4791 | 0.1948 | 9.5744 | 11.3838 | 0.0775 |
| 7 | 10.8621 | 10.8929 | 0.1284 | 10.0252 | 11.7607 | -0.0308 |
| 8 | 11.4083 | 10.8929 | 0.1284 | 10.0252 | 11.7607 | 0.5154 |
| 9 | 10.5419 | 10.8929 | 0.1284 | 10.0252 | 11.7607 | -0.3511 |
| 10 | 11.2988 | 10.8929 | 0.1284 | 10.0252 | 11.7607 | 0.4059 |
| 11 | 10.3294 | 10.8929 | 0.1284 | 10.0252 | 11.7607 | -0.5635 |
| 12 | 10.5328 | 10.8929 | 0.1284 | 10.0252 | 11.7607 | -0.3601 |
| 13 | 10.5899 | 10.9633 | 0.1497 | 10.0852 | 11.8413 | -0.3733 |
| 14 | 10.5752 | 10.9633 | 0.1497 | 10.0852 | 11.8413 | -0.3881 |
| 15 | 11.7530 | 10.9633 | 0.1497 | 10.0852 | 11.8413 | 0.7898 |
| 16 | 11.0174 | 10.9633 | 0.1497 | 10.0852 | 11.8413 | 0.0541 |
| 17 | 11.4140 | 10.9633 | 0.1497 | 10.0852 | 11.8413 | 0.4508 |
| 18 | 10.7584 | 10.9633 | 0.1497 | 10.0852 | 11.8413 | -0.2049 |

Sum of Residuals 0 Sum of Squared Residuals 3.68893 Predicted Residual SS (PRESS) 4.77330

## Dose Proportionality Analysis for Plasma IOXO-292 - AUCO-24 for Figure 14.2.2.8

Model: MODEL1

Dependent Variable: AVAL Analysis Value

Number of Observations Read 18 Number of Observations Used 18

#### Analysis of Variance

| Source | DF | Sum of<br>Squares | Mean<br>Square | F Value | Pr > F |
|---|---|---|---|---|---|
| Model<br>Error<br>Corrected To | 1<br>16<br>tal 17 | 0.87671<br>5.09307<br>5.96979 | 0.87671<br>0.31832 | 2.75 | 0.1165 |
| | Root MSE<br>Dependent Mean<br>Coeff Var | 0.56420<br>10.26685<br>5.49532 | R-Square<br>Adj R-Sq | 0.1469<br>0.0935 | |

# Dose Proportionality Analysis for Plasma LOXO-292 - AUCO-24 for Figure 14.2.2.8

Model: MODEL1

Dependent Variable: AVAL Analysis Value

Parameter Estimates

| Variable | Label | DF | Parameter<br>Estimate | Standard<br>Error | t Value | Pr > t |
|---|---|---|---|---|---|---|
| Intercept | Intercept Log Value of Actual Treatment | 1 | 6.39921 | 2.33428 | 2.74 | 0.0145 |
| LDOSE | | 1 | 0.61688 | 0.37171 | 1.66 | 0.1165 |

## Dose Proportionality Analysis for Plasma IOXO-292 - AUCO-24 for Figure 14.2.2.8

Model: MODEL1 Dependent Variable: AVAL Analysis Value

#### Output Statistics

| Obs | Dependent<br>Variable | Predicted<br>Value | Std Error<br>Mean Predict | 90% CL P | redict | Residual |
|---|---|---|---|---|---|---|
| 1 | 9.8894 | 9.9576 | 0.2289 | 8.8945 | 11.0206 | -0.0681 |
| 2 | 10.6905 | 9.9576 | 0.2289 | 8.8945 | 11.0206 | 0.7329 |
| 3 | 10.5971 | 9.9576 | 0.2289 | 8.8945 | 11.0206 | 0.6396 |
| 4 | 8.9243 | 9.9576 | 0.2289 | 8.8945 | 11.0206 | -1.0333 |
| 5 | 9.3860 | 9.9576 | 0.2289 | 8.8945 | 11.0206 | -0.5716 |
| 6 | 10.3050 | 9.9576 | 0.2289 | 8.8945 | 11.0206 | 0.3474 |
| 7 | 10.3395 | 10.3852 | 0.1509 | 9.3655 | 11.4048 | -0.0456 |
| 8 | 11.0223 | 10.3852 | 0.1509 | 9.3655 | 11.4048 | 0.6371 |
| 9 | 10.0003 | 10.3852 | 0.1509 | 9.3655 | 11.4048 | -0.3848 |
| 10 | 10.7864 | 10.3852 | 0.1509 | 9.3655 | 11.4048 | 0.4012 |
| 11 | 9.8830 | 10.3852 | 0.1509 | 9.3655 | 11.4048 | -0.5022 |
| 12 | 9.9566 | 10.3852 | 0.1509 | 9.3655 | 11.4048 | -0.4286 |
| 13 | 9.9191 | 10.4578 | 0.1759 | 9.4261 | 11.4896 | -0.5387 |
| 14 | 10.0936 | 10.4578 | 0.1759 | 9.4261 | 11.4896 | -0.3642 |
| 15 | 11.3690 | 10.4578 | 0.1759 | 9.4261 | 11.4896 | 0.9112 |
| 16 | 10.5137 | 10.4578 | 0.1759 | 9.4261 | 11.4896 | 0.0559 |
| 17 | 10.8764 | 10.4578 | 0.1759 | 9.4261 | 11.4896 | 0.4186 |
| 18 | 10.2511 | 10.4578 | 0.1759 | 9.4261 | 11.4896 | -0.2067 |

Sum of Residuals 0 Sum of Squared Residuals 5.09307 Predicted Residual SS (PRESS) 6.67982

## Dose Proportionality Analysis for Plasma LOXO-292 - AUCO-inf for Figure 14.2.2.9

Model: MODEL1

Dependent Variable: AVAL Analysis Value

Number of Observations Read 18 Number of Observations Used 18

#### Analysis of Variance

| Source | D | F | Sum of<br>Squares | Mean<br>Square | F Value | Pr > F |
|---|---|---|---|---|---|---|
| Model<br>Error<br>Corrected Tot | | 6 | 0.82655<br>3.69893<br>4.52548 | 0.82655<br>0.23118 | 3.58 | 0.0769 |
| | Root MSE<br>Dependent Mea<br>Coeff Var | n 1 | 0.48082<br>0.78453<br>4.45838 | R-Square<br>Adj R-Sq | 0.1826<br>0.1316 | |

# Dose Proportionality Analysis for Plasma LOXO-292 - AUCO-inf for Figure 14.2.2.9

Model: MODEL1

Dependent Variable: AVAL Analysis Value

Parameter Estimates

| Variable | Label | DF | Parameter<br>Estimate | Standard<br>Error | t Value | Pr > t |
|---|---|---|---|---|---|---|
| Intercept | Intercept Log Value of Actual Treatment | 1 | 7.02918 | 1.98930 | 3.53 | 0.0028 |
| LDOSE | | 1 | 0.59897 | 0.31677 | 1.89 | 0.0769 |

## Dose Proportionality Analysis for Plasma LOXO-292 - AUCO-inf for Figure 14.2.2.9

Model: MODEL1 Dependent Variable: AVAL Analysis Value

#### Output Statistics

| Obs | Dependent<br>Variable | Predicted<br>Value | Std Error<br>Mean Predict | 90% CL | Predict | Residual |
|---|---|---|---|---|---|---|
| 1 | 10.4696 | 10.4842 | 0.1951 | 9.5783 | 11.3902 | -0.0147 |
| 2 | 11.1650 | 10.4842 | 0.1951 | 9.5783 | 11.3902 | 0.6808 |
| 3 | 10.9144 | 10.4842 | 0.1951 | 9.5783 | 11.3902 | 0.4302 |
| 4 | 9.5750 | 10.4842 | 0.1951 | 9.5783 | 11.3902 | -0.9092 |
| 5 | 10.2787 | 10.4842 | 0.1951 | 9.5783 | 11.3902 | -0.2056 |
| 6 | 10.5587 | 10.4842 | 0.1951 | 9.5783 | 11.3902 | 0.0745 |
| 7 | 10.8661 | 10.8994 | 0.1286 | 10.0305 | 11.7684 | -0.0333 |
| 8 | 11.4174 | 10.8994 | 0.1286 | 10.0305 | 11.7684 | 0.5180 |
| 9 | 10.5468 | 10.8994 | 0.1286 | 10.0305 | 11.7684 | -0.3527 |
| 10 | 11.3095 | 10.8994 | 0.1286 | 10.0305 | 11.7684 | 0.4101 |
| 11 | 10.3349 | 10.8994 | 0.1286 | 10.0305 | 11.7684 | -0.5645 |
| 12 | 10.5363 | 10.8994 | 0.1286 | 10.0305 | 11.7684 | -0.3631 |
| 13 | 10.6012 | 10.9700 | 0.1499 | 10.0907 | 11.8492 | -0.3688 |
| 14 | 10.5779 | 10.9700 | 0.1499 | 10.0907 | 11.8492 | -0.3921 |
| 15 | 11.7593 | 10.9700 | 0.1499 | 10.0907 | 11.8492 | 0.7894 |
| 16 | 11.0231 | 10.9700 | 0.1499 | 10.0907 | 11.8492 | 0.0532 |
| 17 | 11.4232 | 10.9700 | 0.1499 | 10.0907 | 11.8492 | 0.4532 |
| 18 | 10.7646 | 10.9700 | 0.1499 | 10.0907 | 11.8492 | -0.2054 |

Sum of Residuals 0
Sum of Squared Residuals 3.69893
Predicted Residual SS (PRESS) 4.78441

# Dose Proportionality Analysis for Plasma IOXO-292 - Cmax for Figure 14.2.2.10

Model: MODEL1

Dependent Variable: AVAL Analysis Value

Number of Observations Read 18 Number of Observations Used 18

#### Analysis of Variance

| Source | | DF | Sum of<br>Squares | Mean<br>Square | F Value | Pr > F |
|---|---|---|---|---|---|---|
| Model<br>Error<br>Corrected To | tal | 1<br>16<br>17 | 0.79125<br>5.61220<br>6.40345 | 0.79125<br>0.35076 | 2.26 | 0.1526 |
| | Root MSE<br>Dependent M<br>Coeff Var | lean | 0.59225<br>8.02245<br>7.38243 | R-Square<br>Adj R-Sq | 0.1236<br>0.0688 | |


# Dose Proportionality Analysis for Plasma IOXO-292 - Cmax for Figure 14.2.2.10

Model: MODEL1

Dependent Variable: AVAL Analysis Value

Parameter Estimates

| Variable | Label | DF | Parameter<br>Estimate | Standard<br>Error | t Value | Pr > t |
|---|---|---|---|---|---|---|
| Intercept | Intercept Log Value of Actual Treatment | 1 | 4.34816 | 2.45036 | 1.77 | 0.0950 |
| LDOSE | | 1 | 0.58604 | 0.39019 | 1.50 | 0.1526 |

# Dose Proportionality Analysis for Plasma IOXO-292 - Cmax for Figure 14.2.2.10

Model: MODEL1 Dependent Variable: AVAL Analysis Value

#### Output Statistics

| Obs | Dependent<br>Variable | Predicted<br>Value | Std Error<br>Mean Predict | 90% CL E | redict | Residual |
|---|---|---|---|---|---|---|
| 1<br>2<br>3<br>4<br>5<br>6<br>7<br>8<br>9<br>10<br>11<br>12<br>13<br>14 | 7.3715<br>8.4764<br>8.4805<br>6.7405<br>7.0901<br>8.2375<br>8.1519<br>8.7499<br>7.8861<br>8.6827<br>7.7187<br>7.4501<br>7.8120<br>7.9725 | 7.7286<br>7.7286<br>7.7286<br>7.7286<br>7.7286<br>7.7286<br>8.1348<br>8.1348<br>8.1348<br>8.1348<br>8.1348<br>8.1348<br>8.2039<br>8.2039 | 0.2403<br>0.2403<br>0.2403<br>0.2403<br>0.2403<br>0.2403<br>0.1584<br>0.1584<br>0.1584<br>0.1584<br>0.1584<br>0.1584<br>0.1584 | 6.6127<br>6.6127<br>6.6127<br>6.6127<br>6.6127<br>7.0645<br>7.0645<br>7.0645<br>7.0645<br>7.0645<br>7.0645<br>7.0645<br>7.1208 | 8.8445<br>8.8445<br>8.8445<br>8.8445<br>8.8445<br>9.2052 | -0.3571<br>0.7477<br>0.7519<br>-0.9881<br>-0.6386<br>0.5088<br>0.0171<br>0.6150<br>-0.2488<br>0.5479<br>-0.4162<br>-0.6848<br>-0.3919<br>-0.2314 |
| 15<br>16<br>17<br>18 | 9.2301<br>8.1017<br>8.2865<br>7.9655 | 8.2039<br>8.2039<br>8.2039<br>8.2039 | 0.1846<br>0.1846<br>0.1846<br>0.1846 | 7.1208<br>7.1208<br>7.1208<br>7.1208 | 9.2869<br>9.2869<br>9.2869<br>9.2869 | 1.0263<br>-0.1022<br>0.0826<br>-0.2383 |

Sum of Residuals 0 Sum of Squared Residuals 5.61220 Predicted Residual SS (PRESS) 7.38988

## **16.1.9.3** Normality Assessments

### Variable: Resid (Residual)

| Moments | | | |
|---|---|---|---|
| N | 18 | Sum Weights | 18 |
| Mean | 0 | <b>Sum Observations</b> | 0 |
| <b>Std Deviation</b> | 0.54735048 | Variance | 0.29959255 |
| Skewness | 0.03401098 | Kurtosis | -0.9501699 |
| <b>Uncorrected SS</b> | 5.09307327 | Corrected SS | 5.09307327 |
| <b>Coeff Variation</b> | | Std Error Mean | 0.12901174 |

| | Basic Statistical Measures | | |
|---|---|---|---|
| Location Variability | | | |
| Mean | 0.00000 | <b>Std Deviation</b> | 0.54735 |
| Median | -0.05687 | Variance | 0.29959 |
| Mode | | Range | 1.94447 |
| | | Interquartile Range | 0.84716 |

| Tests for Location: Mu0=0 | | | | |
|---------------------------|-----------|-----|----------|--------|
| Test | Statistic | | p Value | |
| Student's t | t | 0 | Pr > t | 1.0000 |
| Sign | M | -1 | Pr >= M | 0.8145 |
| Signed Rank | S | 0.5 | Pr >= S | 1.0000 |

| Tests for Normality | | | | |
|---|---|---|---|---|
| Test | Statistic p Value | | | |
| Shapiro-Wilk | W | 0.956817 | Pr < W | 0.5415 |
| Kolmogorov-Smirnov | D | 0.136012 | Pr > D | >0.1500 |
| Cramer-von Mises | W-Sq | 0.058553 | Pr > W-Sq | >0.2500 |
| Anderson-Darling | A-Sq | 0.354958 | Pr > A-Sq | >0.2500 |

| Quantiles (D | Definition 5) |
|--------------|---------------|
| Quantile | Estimate |
| 100% Max | 0.911191 |
| 99% | 0.911191 |
| 95% | 0.911191 |
| 90% | 0.732887 |
| 75% Q3 | 0.418596 |
| 50% Median | -0.056869 |
| 25% Q1 | -0.428560 |
| 10% | -0.571557 |
| 5% | -1.033276 |
| 1% | -1.033276 |
| 0% Min | -1.033276 |

| <b>Extreme Observations</b> | | | |
|-----------------------------|-----|----------|-----|
| Lowes | t | Highest | |
| Value | Obs | Value | Obs |
| -1.033276 | 4 | 0.418596 | 17 |
| -0.571557 | 5 | 0.637136 | 8 |
| -0.538749 | 13 | 0.639577 | 3 |
| -0.502206 | 11 | 0.732887 | 2 |
| -0.428560 | 12 | 0.911191 | 15 |





### Fitted Normal Distribution for Resid (Residual)

| Parameters for Normal<br>Distribution | | |
|---------------------------------------|-------|---------|
| Parameter Symbol Estimate | | |
| Mean | Mu | 0 |
| Std Dev | Sigma | 0.54735 |

| Goodness-of-Fit Tests for Normal Distribution | | | | |
|---|---|---|---|---|
| Test | Statistic p Value | | | |
| Kolmogorov-Smirnov | D | 0.13601194 | Pr > D | >0.150 |
| Cramer-von Mises | W-Sq | 0.05855315 | Pr > W-Sq | >0.250 |
| Anderson-Darling | A-Sq | 0.35495841 | Pr > A-Sq | >0.250 |

| Quantiles for Normal Distribution | | |
|-----------------------------------|----------|-----------|
| | Quantile | |
| Percent | Observed | Estimated |
| 1.0 | -1.03328 | -1.27333 |
| 5.0 | -1.03328 | -0.90031 |
| 10.0 | -0.57156 | -0.70146 |
| 25.0 | -0.42856 | -0.36918 |
| 50.0 | -0.05687 | 0.00000 |
| 75.0 | 0.41860 | 0.36918 |
| 90.0 | 0.73289 | 0.70146 |
| 95.0 | 0.91119 | 0.90031 |
| 99.0 | 0.91119 | 1.27333 |



### Variable: Resid (Residual)

| | Moments | | |
|---|---|---|---|
| N | 18 | Sum Weights | 18 |
| Mean | 0 | <b>Sum Observations</b> | 0 |
| <b>Std Deviation</b> | 0.46582814 | Variance | 0.21699586 |
| Skewness | 0.02529015 | Kurtosis | -0.7048472 |
| <b>Uncorrected SS</b> | 3.68892959 | Corrected SS | 3.68892959 |
| <b>Coeff Variation</b> | | Std Error Mean | 0.10979675 |

| | Basic Statistical Measures | | |
|---|---|---|---|
| Location Variability | | | |
| Mean | 0.00000 | <b>Std Deviation</b> | 0.46583 |
| Median | -0.02241 | Variance | 0.21700 |
| Mode | • | Range | 1.69726 |
| | | Interquartile Range | 0.79460 |

| Tests for Location: Mu0=0 | | | | |
|---------------------------|-------------------|-----|----------|--------|
| Test | Statistic p Value | | | ue |
| Student's t | t | 0 | Pr > t | 1.0000 |
| Sign | M | -1 | Pr >= M | 0.8145 |
| Signed Rank | S | 4.5 | Pr >= S | 0.8650 |

| Tests for Normality | | | | |
|---------------------|------|-----------------|-----------|---------|
| Test | Sta | Statistic p Val | | |
| Shapiro-Wilk | W | 0.963641 | Pr < W | 0.6731 |
| Kolmogorov-Smirnov | D | 0.14155 | Pr > D | >0.1500 |
| Cramer-von Mises | W-Sq | 0.05408 | Pr > W-Sq | >0.2500 |
| Anderson-Darling | A-Sq | 0.323198 | Pr > A-Sq | >0.2500 |

| <b>Quantiles (Definition 5)</b> | |
|---------------------------------|------------|
| Quantile | Estimate |
| 100% Max | 0.7897647 |
| 99% | 0.7897647 |
| 95% | 0.7897647 |
| 90% | 0.6790547 |
| 75% Q3 | 0.4344805 |
| 50% Median | -0.0224074 |
| 25% Q1 | -0.3601238 |
| 10% | -0.5634883 |
| 5% | -0.9074926 |
| 1% | -0.9074926 |
| 0% Min | -0.9074926 |

| <b>Extreme Observations</b> | | | |
|-----------------------------|--------|----------|-----|
| Lowes | Lowest | | est |
| Value | Obs | Value | Obs |
| -0.907493 | 4 | 0.434481 | 3 |
| -0.563488 | 11 | 0.450776 | 17 |
| -0.388061 | 14 | 0.515411 | 8 |
| -0.373340 | 13 | 0.679055 | 2 |
| -0.360124 | 12 | 0.789765 | 15 |





### Fitted Normal Distribution for Resid (Residual)

| Parameters for Normal<br>Distribution | | |
|---------------------------------------|-------|----------|
| Parameter Symbol Estimate | | |
| Mean | Mu | 0 |
| Std Dev | Sigma | 0.465828 |

| Goodness-of-Fit Tests for Normal Distribution | | | | |
|---|---|---|---|---|
| Test | Statistic p Value | | | ie |
| Kolmogorov-Smirnov | D | 0.14154968 | Pr > D | >0.150 |
| Cramer-von Mises | W-Sq | 0.05408010 | Pr > W-Sq | >0.250 |
| Anderson-Darling | A-Sq | 0.32319805 | Pr > A-Sq | >0.250 |

| Quantiles for Normal<br>Distribution | | |
|--------------------------------------|----------|-----------|
| | Quantile | |
| Percent | Observed | Estimated |
| 1.0 | -0.90749 | -1.08368 |
| 5.0 | -0.90749 | -0.76622 |
| 10.0 | -0.56349 | -0.59698 |
| 25.0 | -0.36012 | -0.31420 |
| 50.0 | -0.02241 | 0.00000 |
| 75.0 | 0.43448 | 0.31420 |
| 90.0 | 0.67905 | 0.59698 |
| 95.0 | 0.78976 | 0.76622 |
| 99.0 | 0.78976 | 1.08368 |



### Variable: Resid (Residual)

| Moments | | | |
|---|---|---|---|
| N | 18 | 8 Sum Weights | |
| Mean | 0 | <b>Sum Observations</b> | 0 |
| <b>Std Deviation</b> | 0.46645909 | Variance | 0.21758408 |
| Skewness | 0.02449645 | Kurtosis | -0.7030042 |
| <b>Uncorrected SS</b> | 3.69892938 | Corrected SS | 3.69892938 |
| <b>Coeff Variation</b> | | Std Error Mean | 0.10994546 |

| Basic Statistical Measures | | | |
|---|---|---|---|
| Loca | Location Variability | | |
| Mean | 0.00000 | <b>Std Deviation</b> | 0.46646 |
| Median | -0.02399 | Variance | 0.21758 |
| Mode | | Range | 1.69857 |
| | | Interquartile Range | 0.79328 |

| Tests for Location: Mu0=0 | | | | |
|---------------------------|-------------------|-----|----------|--------|
| Test | Statistic p Value | | | |
| Student's t | <b>t</b> 0 | | Pr > t | 1.0000 |
| Sign | M | -1 | Pr >= M | 0.8145 |
| Signed Rank | S | 4.5 | Pr >= S | 0.8650 |

| Tests for Normality | | | | |
|---|---|---|---|---|
| Test | Statistic p Value | | | |
| Shapiro-Wilk | W | 0.963429 | Pr < W | 0.6689 |
| Kolmogorov-Smirnov | D | 0.143674 | Pr > D | >0.1500 |
| <b>Cramer-von Mises</b> | W-Sq | 0.054387 | Pr > W-Sq | >0.2500 |
| Anderson-Darling | A-Sq | 0.324758 | Pr > A-Sq | >0.2500 |

| <b>Quantiles (Definition 5)</b> | |
|---------------------------------|------------|
| Quantile | Estimate |
| 100% Max | 0.7893745 |
| 99% | 0.7893745 |
| 95% | 0.7893745 |
| 90% | 0.6807874 |
| 75% Q3 | 0.4301697 |
| 50% Median | -0.0239911 |
| 25% Q1 | -0.3631091 |
| 10% | -0.5645001 |
| 5% | -0.9091996 |
| 1% | -0.9091996 |
| 0% Min | -0.9091996 |

| <b>Extreme Observations</b> | | | |
|-----------------------------|----|----------|-----|
| Lowes | t | Highe | est |
| Value Obs | | Value | Obs |
| -0.909200 | 4 | 0.430170 | 3 |
| -0.564500 | 11 | 0.453220 | 17 |
| -0.392096 | 14 | 0.517990 | 8 |
| -0.368800 | 13 | 0.680787 | 2 |
| -0.363109 | 12 | 0.789374 | 15 |





### Fitted Normal Distribution for Resid (Residual)

| Parameters for Normal<br>Distribution | | |
|---------------------------------------|-------|----------|
| Parameter Symbol Estimate | | |
| Mean | Mu | 0 |
| Std Dev | Sigma | 0.466459 |

| Goodness-of-Fit Tests for Normal Distribution | | | | |
|---|---|---|---|---|
| Test | Statistic p Value | | | |
| Kolmogorov-Smirnov | D | 0.14367408 | Pr > D | >0.150 |
| Cramer-von Mises | W-Sq | 0.05438651 | Pr > W-Sq | >0.250 |
| Anderson-Darling | A-Sq | 0.32475804 | Pr > A-Sq | >0.250 |

| Quantiles for Normal<br>Distribution | | |
|--------------------------------------|----------|-----------|
| | Quantile | |
| Percent | Observed | Estimated |
| 1.0 | -0.90920 | -1.08515 |
| 5.0 | -0.90920 | -0.76726 |
| 10.0 | -0.56450 | -0.59779 |
| 25.0 | -0.36311 | -0.31462 |
| 50.0 | -0.02399 | 0.00000 |
| 75.0 | 0.43017 | 0.31462 |
| 90.0 | 0.68079 | 0.59779 |
| 95.0 | 0.78937 | 0.76726 |
| 99.0 | 0.78937 | 1.08515 |



### Variable: Resid (Residual)

| Moments | | | |
|---|---|---|---|
| N | 18 | 18 Sum Weights | |
| Mean | 0 | <b>Sum Observations</b> | 0 |
| <b>Std Deviation</b> | 0.57456894 | Variance | 0.33012946 |
| Skewness | 0.23968228 | Kurtosis | -0.950472 |
| <b>Uncorrected SS</b> | 5.61220085 | Corrected SS | 5.61220085 |
| <b>Coeff Variation</b> | | Std Error Mean | 0.1354272 |

| Basic Statistical Measures | | | |
|----------------------------|----------|----------------------|---------|
| Location Variability | | | |
| Mean | 0.00000 | <b>Std Deviation</b> | 0.57457 |
| Median | -0.16680 | Variance | 0.33013 |
| Mode | | Range | 2.01438 |
| | | Interquartile Range | 0.93976 |

| Tests for Location: Mu0=0 | | | | |
|---------------------------|-------------------|------|----------|--------|
| Test | Statistic p Value | | | |
| Student's t | t | 0 | Pr > t | 1.0000 |
| Sign | M | -1 | Pr >= M | 0.8145 |
| Signed Rank | S | -0.5 | Pr >= S | 1.0000 |

| Tests for Normality | | | | |
|---------------------|-----------|----------|-----------|---------|
| Test | Statistic | | p Value | |
| Shapiro-Wilk | W | 0.950454 | Pr < W | 0.4322 |
| Kolmogorov-Smirnov | D | 0.156434 | Pr > D | >0.1500 |
| Cramer-von Mises | W-Sq | 0.078884 | Pr > W-Sq | 0.2084 |
| Anderson-Darling | A-Sq | 0.433324 | Pr > A-Sq | >0.2500 |

| <b>Quantiles (Definition 5)</b> | |
|---------------------------------|-----------|
| Quantile | Estimate |
| 100% Max | 1.026269 |
| 99% | 1.026269 |
| 95% | 1.026269 |
| 90% | 0.751894 |
| 75% Q3 | 0.547859 |
| 50% Median | -0.166802 |
| 25% Q1 | -0.391901 |
| 10% | -0.684769 |
| 5% | -0.988116 |
| 1% | -0.988116 |
| 0% Min | -0.988116 |

| <b>Extreme Observations</b> | | | |
|-----------------------------|-----|----------|-----|
| Lowest | | Highest | |
| Value | Obs | Value | Obs |
| -0.988116 | 4 | 0.547859 | 10 |
| -0.684769 | 12 | 0.615043 | 8 |
| -0.638559 | 5 | 0.747736 | 2 |
| -0.416163 | 11 | 0.751894 | 3 |
| -0.391901 | 13 | 1.026269 | 15 |





### Fitted Normal Distribution for Resid (Residual)

| Parameters for Normal<br>Distribution | | |
|---------------------------------------|--------|----------|
| Parameter | Symbol | Estimate |
| Mean | Mu | 0 |
| Std Dev | Sigma | 0.574569 |

| Goodness-of-Fit Tests for Normal Distribution | | | | |
|---|---|---|---|---|
| Test | Statistic | | p Value | |
| Kolmogorov-Smirnov | D | 0.15643424 | Pr > D | >0.150 |
| Cramer-von Mises | W-Sq | 0.07888421 | Pr > W-Sq | 0.208 |
| Anderson-Darling | A-Sq | 0.43332377 | Pr > A-Sq | >0.250 |

| Quantiles for Normal<br>Distribution | | |
|--------------------------------------|----------|-----------|
| | Quantile | |
| Percent | Observed | Estimated |
| 1.0 | -0.98812 | -1.33665 |
| 5.0 | -0.98812 | -0.94508 |
| 10.0 | -0.68477 | -0.73634 |
| 25.0 | -0.39190 | -0.38754 |
| 50.0 | -0.16680 | 0.00000 |
| 75.0 | 0.54786 | 0.38754 |
| 90.0 | 0.75189 | 0.73634 |
| 95.0 | 1.02627 | 0.94508 |
| 99.0 | 1.02627 | 1.33665 |

